

# **Non-interventional Study Protocol**

| Document Number: | c25576073-03 |
|---|---|
| BI Study Number: | 1199-0355 |
| BI Investigational | Ofev®, nintedanib |
| Product(s): | |
| Title: | Investigating Trends in Quality of Life in Patients with |
| | Idiopathic Pulmonary Fibrosis (IPF) Under Treatment |
| | with Nintedanib |
| Brief lay title | QUALIFY Idiopathic Pulmonary Fibrosis |
| <b>Protocol version</b> | 3.0 |
| identifier: | |
| Date of last version of | 11 February 2021 |
| protocol: | |
| PASS: | No |
| EU PAS register | Not yet registered |
| number: | |
| Active substance: | Pharmacotherapeutic group: Antineoplastic agents, |
| | protein kinase inhibitors, ATC code: L01XE31 |
| Medicinal product: | OFEV,100 mg and 150 mg soft capsules |
| Product reference: | EU/1/14/979 |
| Procedure number: | EMEA/H/C/3821/WS/1307 |
| Marketing authorization | Boehringer Ingelheim International GmbH |
| holder(s): | |

| Joint PASS: | No |
|---|---|
| Research question and objectives: | The aim of this non-interventional-study is to collect data on various important Patient Reported Outcomes (PROs) in patients with IPF that could provide useful insights about Health-Related Quality of Life (HRQoL) over 52 weeks in patients treated with nintedanib in the real world setting in Greece. Primary objective: - To evaluate HRQoL changes from baseline for IPF patients treated in current clinical practice in Greece with nintedanib at time-points of 3, 6, 9 and 12 months over a 52-week period, via SGRQ. |
| | <ul> <li>Secondary objectives are:</li> <li>To assess changes, from baseline, in dyspnoea and cough in IPF patients treated with nintedanib in current clinical practice in Greece at time-points of 3, 6, 9 and 12 months over a 52 weeks period, via specific questionnaires, such as mMRC score and Cough - Visual Analogue Scale (Cough - VAS) respectively.</li> <li>To evaluate the adherence to nintedanib treatment in current clinical practice at time-points of 3, 6, 9 and 12 months over a 52 weeks period via SMAQ Questionnaire (adapted for the treatment of idiopathic pulmonary fibrosis (IPF).</li> <li>To measure anxiety in IPF patients treated with nintedanib in current clinical practice in Greece at time-points of baseline, 3, 6, 9 and 12 months over a 52 weeks period via GAD-7 Questionnaire.</li> </ul> |

| | - To estimate the use of Long-Term Oxygen Treatment (LTOT) among IPF patients under treatment with nintedanib in current clinical practice in Greece at timepoints of baseline, 3, 6, 9 and 12 months over a 52 weeks period. |
|---|---|
| Country(-ies) of study: | Greece |
| Author: | |
| Marketing authorisation holder(s): | Boehringer Ingelheim |
| In case of PASS, add: MAH contact person: | Not applicable |
| In case of PASS, add: <eu-qppv:></eu-qppv:> | Not applicable |
| In case of PASS, add: <signature eu-="" of="" qppv:=""></signature> | Not applicable |
| Date: | 11 February 2021 |
| Page 3 of 104 | |

# **Proprietary confidential information**

# © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

# 1. TABLE OF CONTENTS

| TITLE P | 'AGE | 1 |
|---|---|---|
| 1. T | ABLE OF CONTENTS | 4 |
| 2. L | IST OF ABBREVIATIONS | 6 |
| | RESPONSIBLE PARTIES | Q |
| 4. A | ABSTRACT | |
| | Nintedanib treatment (start date, dose) | |
| | Assessment of lung function and exercise capacity (FVC, DLCO, 6-minutes walking test) | |
| | <ul> <li>Physical and vital signs examination (blood pressure, heart rate)</li> <li>Nintedanib treatment (stop date, restart date in case of temporary discontinuation, dose)</li> </ul> | |
| 5. A | AMENDMENTS AND UPDATES | 31 |
| 6. N | MILESTONES | 39 |
| 7. R | RATIONALE AND BACKGROUND | 40 |
| | DEFINITION | |
| 7.1 | INCIDENCE AND PREVALENCE | |
| 7.2<br>7.3 | DIAGNOSIS | |
| 7.3 | NATURAL COURSE | |
| 7.5 | THERAPY | |
| 7.6 | RATIONALE FOR THE PRESENT STUDY | |
| 7.6.1 | | |
| 8. R | RESEARCH QUESTION AND OBJECTIVES | 46 |
| | RESEARCH METHODS | |
| 9.1 | STUDY DESIGN | |
| 9.1 | SETTING | |
| 9.2.1 | | |
| 9.2.2 | | |
| 9.2.3 | | |
| 9.2.4 | Patient discontinuation | 49 |
| 9.2.5 | , | |
| 9.3 | VARIABLES | |
| 9.3.1 | ! | |
| 9.3.2 | · · | |
| | 9.3.2.1 Primary endpoint | |
| | 3.3.2.2 Secondary endpoints | |
| 9.3.3 | Covariates | 53 |
| 9.4 | DATA SOURCES | 57 |
| 9.5 | STUDY SIZE | 59 |
| 9.6 | DATA MANAGEMENT | |
| 9.7 | DATA ANALYSIS | |
| 9.7.1 | Main analysis | 62 |
| 0.0 | OLIALITY CONTROL | |
| 9.8 | QUALITY CONTROL | 63<br>64 |

| 9.10 | OTHER ASPECTS | 65 |
|---|---|---|
| 9.10.1 | Data quality assurance | 65 |
| 9.10.2 | Study records | 66 |
| | 9.10.2.1 Source documents | |
| | 9.10.2.2 Direct access to source data and documents | |
| | 9.10.2.3 Storage of records | |
| 9.10.3 | Completion of study | <i>6</i> 8 |
| 10. PF | OTECTION OF HUMAN SUBJECTS | 69 |
| 10.1 | STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT | 69 |
| | STATEMENT OF CONFIDENTIALITY | |
| 11. M | ANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 72 |
| | DEFINITIONS OF ADVERSE EVENTS | |
| 11.2 | ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING | 73 |
| 11.3 | REPORTING TO HEALTH AUTHORITIES | 77 |
| 12. PL | ANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 78 |
| 13. RE | FERENCES | 80 |
| 13.1 | PUBLISHED REFERENCES | 80 |
| 13.2 | UNPUBLISHED REFERENCES | 82 |
| ANNEX : | . LIST OF STAND-ALONE DOCUMENTS | 83 |
| ANNEX | 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 84 |
| ANNEX | 3. ADDITIONAL INFORMATION | 94 |

### 2. LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event

AESI Adverse Event of Special interest

ALAT Latin American Thoracic Association

ATS American Thoracic Society

CA Competent Authority

CCDS Company Core Data Sheet

CI Confidence Interval

CRA Clinical Research Associate

CRF Case Report Form

CRO Clinical Research Organization

CTCAE Common Terminology Criteria for Adverse Events

CTM Clinical Trial Manager
CTP Clinical Trial Protocol
DMP Data Management Plan

eCRF Electronic Case Report Form

ENCePP European Network of Centres for Pharmacoepidemiology and

PV Pharmacovigilance

ERS European Respiratory Society
FDA Food and Drug Administration

FGF Fibroblast Growth Factor

FVC Forced Vital Capacity

GAD-7 Generalized Anxiety Disorder Screener Questionnaire

GCP Good Clinical Practice

GEP Good Epidemiological Practice

GPP Good Pharmacoepidemiology Practice
GVP Good Pharmacovigilance Practices

HRCT High Resolution Computer Tomography

HRQoL Health Related Quality of Life

IB Investigator's Brochure

IEC Independent Ethics CommitteeIIP Idiopathic Interstitial Pneumonia

ILD Interstitial Lung Disease

IPF Idiopathic Pulmonary Fibrosis
IRB Institutional Review Board
JRS Japanese Respiratory Society
LTOT Long Term Oxygen Therapy

MAH Marketing Authorization Holder

mMRC modified Medical Research Council scale

NIS Non-Interventional Study

PASS Post-Authorization Safety Study
PDGF Platelet Derived Growth Factor

PROs Patient Reported Outcomes
RCT Randomized Clinical Trial

SAE Serious Adverse Event SAP Statistical Analysis Plan

SD Standard Deviation

SGRQ St. George's Respiratory Questionnaire

SMAQ Simplified Medication Adherence Questionnaire

SmPC Summary of Product Characteristics

UIP Usual Interstitial Pneumonia

VAS Visual Analogue Scale

VEGF Vascular Endothelial Growth Factor

# 3. RESPONSIBLE PARTIES

**Trial Sponsor** 



# **Participating Investigators**

A contact list of the participating investigators will be stored as a standalone (independent) document and will be available upon request.

# 4. ABSTRACT

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingel | heim | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| Protocol date: | Study | Version/Revision: 3.0 | Version/Revision date: |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Rationale and | IPF is a rare, c | hronic and progressive pulmona | ry disease affecting 2.8-9.3 |
| background: | persons per 1 | 00,000 in the western world ( | 1). IPF is associated with |
| | chronic dyspn | oea and cough and the progres | sive loss of lung function, |
| leading to resp | | piratory failure (2). However, th | e clinical course of disease |
| | is variable with some patients progressing slowly, others rapidly and | | |
| | some patients | experiencing acute exacerbatio | ns that are associated with |
| | increased mo | rbidity and mortality (3). Ur | ntil recently no effective |
| | pharmacological treatment besides lung transplantation was available for | | |
| | IPF patients. Nintedanib, an oral multi-tyrosine kinase inhibitor, was | | |
| | approved in EU on January 2015 for the treatment of IPF patients | | |
| | independent of the stage of their disease (4). Nintedanib is available and | | |
| | reimbursed in Greece since February 2016. Due to the rarity of IPF, there | | |
| | | ed data regarding the patients' population, the natural course | |
| | of the disease and the medical treatment these patients receive, as | | |
| | highlighted by | the call for action towards a wo | orldwide IPF registry (5). |

| Name of compan | ny: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating Trends in Quality of Life in Patients with IPF Under | | ients with IPF Under |
| | Treatment with Nintedanib | | |
| Rationale and | Especially for the Greek population, very few data are available | | |
| background | regarding the | use of nintedanib in cohorts of p | patients with IPF either pre- |
| (cont'd): | treated or trea | atment-naïve, also in terms of Pa | atients Reported Outcomes |
| | (PRO) (6). T | he recently launched observation | onal study INDULGE-IPF |
| | (NCT030741 | 49) will provide essential data re | egarding the natural course |
| | of IPF and the treatment of the disease – including the use of nintedanib | | |
| | – in the Gree | ek population. In a chronic dis | ease like IPF, the goal of |
| | pharmacological treatments should not be only survival prolongation, | | |
| | but also delay in the progression of the disease and on the clinical | | |
| | deterioration of patients, i.e. delay worsening of symptoms and quality | | |
| | of life. In IPF, there is a paucity of well validated PRO measures. In the | | |
| | pooled analysis of nintedanib randomized trials in IPF, the use of SGRQ | | |
| | questionnaire as a measurement of health related quality of life provided | | |
| | evidence for a modest effect of nintedanib on the delay of clinical | | |
| | deterioration | of patients (4, 7). | |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Patients with IPF Under | |
| | Treatment wi | th Nintedanib | |
| Rationale and | In addition a | a German IPF registry (INS) | IGHTS-IPF) has recently |
| background | published res | ults for patient reported outc | omes (PROs) in enrolled |
| (cont'd): | patients, show | ving IPF patients under real-l | ife conditions have lower |
| | HRQoL compared to those in clinical studies (8). In the Greek population, | | 8). In the Greek population, |
| | analogous results regarding the effect of nintedanib on SGRQ as well as | | |
| | other PRO measures are lacking. Therefore, the aim of this non- | | |
| | interventional-study based on newly collected data is to collect data on | | |
| | various important PROs in patients with IPF that could provide useful | | |
| | insights about HRQoL over 52 weeks in patients treated with nintedanib | | |
| | in the real wor | rld setting in Greece. | |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingel | heim | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating Trends in Quality of Life in Patients with IPF Under | | |
| | Treatment with Nintedanib | | |
| Research | Primary objective: | | |
| question and | - To evaluate the HRQoL changes of IPF patients treated in current | | |
| objectives: | clinical pr | actice in Greece with nintedan | ib at time-points of 3, 6, 9 |
| | and 12 months over a 52-weeks period, via SGRQ. | | |
| | Secondary objectives are: | | |
| | - To assess changes, from baseline, in dyspnoea and cough in IPF | | |
| | patients treated with nintedanib in current clinical practice in Greece | | |
| | at time-points of 3, 6, 9 and 12 months over a 52 weeks period, via | | |
| | specific qu | uestionnaires, such as mMRC so | ore and Cough – Visual |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Research | Analogue Scale (Cough - VAS) respectively. | | ly. |
| question and | - To evaluate the adherence to nintedanib treatment in current clinical | | reatment in current clinical |
| objectives | practice at | time-points of 3, 6, 9 and 12 mor | nths over a 52 weeks period |
| (cont'd): | via SMAQ | Questionnaire (adapted for the | ne treatment of idiopathic |
| | pulmonary fibrosis (IPF). | | |
| | - To measure anxiety in IPF patients treated with nintedanib in current | | |
| | clinical practice in Greece at time-points of baseline, 3, 6, 9 and 12 | | |
| | months over a 52 weeks period via GAD-7 Questionnaire. | | |
| | - To estimate the use of Long-Term Oxygen Treatment (LTOT) among | | |
| | IPF patient | ts under treatment with nintedani | b in current clinical practice |
| | in Greece | at time-points of baseline, 3, 6, | 9 and 12 months over a 52 |
| | weeks peri | od. | |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Study design: | This is a Nati | onal, multi-center, non-interver | ntional, prospective cohort |
| | study aiming | g to enroll 240 IPF patients | receiving treatment with |
| | nintedanib in a consecutive manner from 10-12 reference centers across | | |
| | Greece, representative of the entire Greek population. Recruitment will | | |
| | last for 36 months and patients will be followed over a period of 52 | | |
| | weeks. A baseline visit and 4 follow up visits will be performed during | | |
| | the follow-up | period according to clinical pra | ctice. |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingel | heim | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | - |
| ATC code: L01X | Œ31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Study design | In the context | of this study, participating ph | ysicians shall follow each |
| (cont'd): enrolled patien | | nt for a planned observation per | riod of 12 months, starting |
| | from the date | of baseline visit and ending a | t the earliest of treatment |
| | discontinuation | n, withdrawal of consent, physic | eian's decision to withdraw |
| the patient, 12 | | -month observation period com | pletion, death or any other |
| | discontinuation | n criterion is met. | |
| | Patients that w | rithdraw from the study (consent | withdrawal, lost to Follow |
| | up) or permanently discontinue nintedanib treatment, prior to the follow | | |
| | up period completion, for any reason (e.g. due to AE, physician's | | |
| | decision), will no longer be followed-up for the study and the visit that | | |
| | discontinuation is recorded will be considered as their end of study visit. | | |
| | Patients that temporarily interrupt treatment with nintedanib, up to 28 | | |
| days, will continue f | | tinue follow up activities accor | ding to the study plan and |
| | will not be dis | continued from the study. | |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | - |
| ATC code: L01X | Œ31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Par | tients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Population: | In this study, | there will be enrolled approxin | nately 240 consecutive IPF |
| | patients from 10-12 sites – Academic Hospitals and reference centres. | | |
| | Participating centres and therefore participating physicians have large | | |
| | experience in the management of patients with IPF and may also be part | | |
| | of a larger referral network. | | |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingel | heim | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | |
| ATC code: L01X | Œ31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Population | Patients will b | be eligible to enrol in the study is | f they fulfil all the inclusion |
| (cont'd): | criteria and no | one of the exclusion criteria: | |
| | Inclusion crite | <u>ria</u> | |
| | • Patients ≥ | 240 years of age. | |
| | Patients tl | hat have signed Informed Conse | nt Form. |
| | Treatmen | t naïve patients with an initial I | PF diagnosis no more than |
| | 3 months | prior to enrolment according to 2 | 2011 ATS/ERS/JRS/ALAT |
| | guideline | s and have initiated treatme | ent with Nintedanib (as |
| | monother | apy for IPF) within the past 7 day | ys prior to study enrolment. |
| | • Patients f | or whom the decision to prescri | be therapy with nintedanib |
| | according to the locally approved product's Summary of Product | | |
| | Characteristics (SmPC) has already been taken prior to their | | |
| | enrolment in the study and is clearly separated from the physici | | |
| | decision to include the patient in the current study. | | |
| | Patients that are able to read, understand and complete the study | | |
| | specific q | uestionnaires. | |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Population | Exclusion | <u>criteria</u> | |
| (cont'd): | Treatment with nintedanib for more than 7 days prior to study | | |
| | enrolment. | | |
| | Patients receiving a combination therapy of nintedanib & pirfenidone | | |
| | for IPF. | | |
| | • Patients th | nat meet any of the contraindica | ations to the administration |
| | of the study drug nintedanib according to the approved SmPC. | | |
| | Prior treatment with pirfenidone or other treatment for IPF. | | |
| | Patients participate in an interventional trial, currently receiving | | |
| | treatment with any investigational drug/device/intervention or | | |
| | having received any investigational product within 1 month or 5 half- | | |
| | lives of t | of the investigational agent (whichever is longer) before the | |
| | initiation | of therapy with nintedanib. | |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingel | heim | | |
| Name of finished medicinal | | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | |
| ATC code: L01X | Œ31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| | status of IPF p Basic ( Anthro Physica rate) IPF rish Co-mod categor Record IPF and IPF syr Ninteda Assessi | relevant patient history will be reatients will be recorded regarding Socio-) demographic data pometric characteristics (body was all and vital signs examination (as k factors residities and concomitant ry/class) ling of the methods and procedured date of diagnosis (including Himptoms anib treatment (start date, dose) ment of lung function and exercites walking test) | veight, height) reterial/blood pressure, heart treatments (medication res used in the diagnosis of RCT and SLB) |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment with Nintedanib | | |
| Variables | Questionnaires (SGRQ, mMRC Score, Cough - VAS, GAD-7 ) | | |
| (cont'd): | Long Term Oxygen Therapy | | |
| | The following variables will be also recorded at follow up visits: | | |
| | • Physica | al and vital signs examination (b | lood pressure, heart rate) |
| | • Anthro | pometric characteristics (body w | veight) |
| | Nintedanib treatment (stop date, restart date in case of temporary) | | |
| | discontinuation, dose) | | |
| | Questionnaires (SGRQ, mMRC Score, Cough - VAS, SMAQ, | | |
| | GAD-7) | | |
| | Long Term Oxygen Therapy | | |
| | Changes in concomitant treatments (medication category/class). | | |
| | • Surviva | al status | |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment with Nintedanib | | |
| Data sources: | New data co | ollection. Data will be recorde | ed via e-CRF, where the |
| | participating | physician will record both clin | ical data, such as baseline |
| | characteristics and other medical data, and also the data from the relevant | | |
| | questionnaires that the patient will have to fill out either alone or in | | |
| | collaboration with the participating physician or the study nurse, if | | |
| | available. The following questionnaires will be used for this study: | | |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pa | ntients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Data sources | -SGRQ is a | self-administered, 50-item qu | estionnaire assessing three |
| (cont'd): | domains: s | symptoms, activity and impact. | This questionnaire has been |
| | validated f | for use in patients with COPD | but also has been tested for |
| | patients w | ith IPF and could detect alterat | tions in the clinical status of |
| | the patient | s. The total score and the score | for each domain range from |
| | 0 to 100, v | with higher scores indicating wo | orse health-related quality of |
| | life. A mi | inimally important difference | in the score has not been |
| | established | d for patients with idiopathic pu | llmonary fibrosis; in patients |
| | with chro | nic obstructive pulmonary di | sease, this difference is 4 |
| | points. | | |
| | -mMRC is a modified medical research council dyspnoea scale that uses | | |
| | same descriptors as the original MRC scale. The descriptors of the | | |
| | mMRC scale are numbered 1-5 and are used to estimate the patient's | | |
| | perception of breathlessness. The specific scale has been validated as | | |
| | a measurer | ment of disease severity in IPF | patients. |

| Boehringer Ingell | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pati | ients with IPF Under |
| | Treatment wi | Treatment with Nintedanib | |
| Data sources | -Cough - VAS is recommended as an instrument for the assessment of | | |
| (cont'd): | IPF related cough. | | |
| | -SMAQ is a validated six-item questionnaire that estimates in a | | |
| | qualitative | and semi-quantitative manner the | he adherence of patients to |
| | treatment. | | |
| | - GAD-7 is a 7-item instrument validated for anxiety evaluation that could | | |
| | be used in outpatient setting. | | |
| | All questionnaires should be administered to the patients for | | |
| | completion at the beginning of their visit by the treating physician and | | |
| | prior to any clinical evaluation. All these completed questionnaires | | |
| | will be stored safely in the centres for future purposes of Data Review | | |
| | & Quality | Checks if needed. | |
| Title of study: Data sources | Investigating Treatment wi -Cough - VAS IPF related -SMAQ is a qualitative treatmentGAD-7 is a 7 be used in All questi completion prior to an will be store | S is recommended as an instrument cough. I validated six-item questions and semi-quantitative manner the item instrument validated for an outpatient setting. I ionnaires should be administed at the beginning of their visit by any clinical evaluation. All these red safely in the centres for future | nent for the assessment aire that estimates in the adherence of patients existing evaluation that con- |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | neim | | |
| Name of finished medicinal | | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Primary and | The primary | endpoint of the study is: | |
| Secondary | • The m | ean change from baseline in H | IRQoL (with reference to |
| Endpoints | SGRQ score, both total score and score of each of the SGRQ | | |
| | domain) in patients under treatment with nintedanib, as assessed | | |
| | at time | -point3, 6, 9 and 12 months over | er the 52 weeks follow-up |
| | period. | | |
| | The secondary | endpoints of the study are: | |
| | • Change | e from baseline to 3, 6, 9 and 12 | 2 months follow up period |
| | of dysp | onoea burden as measured by mM | MRC score at time-point |
| | • The mean change from baseline to 3, 6, 9 and 12 months follow | | |
| | up period of cough burden, as measured via changes in the Cough | | |
| | - Visual Analogue Scale (cough - VAS) for coughtime-point | | |
| | Percentage of adhered patients to nintedanib treatment at time- | | |
| | points | points of 3, 6, 9 and 12 months over the 52 weeks follow up period, | |
| | as measured via SMAQ questionnaire (adapted for the treatment | | |
| | of idio | pathic pulmonary fibrosis (IPF). | |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of finished | d medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | - |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Par | tients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Primary and | • The me | ean change from baseline to 3, | 6, 9 and 12 months follow |
| Secondary | up period of anxiety in patients treated with nintedanib at time- | | |
| Endpoints | point as measured via GAD-7 questionnaire. | | |
| (cont'd): | • Percentage of patients that use LTOT at time-points of 3, 6, 9 and | | |
| | 12 months over the 52 weeks follow up period. | | |
| Study size: | This observational study will be analyzed using descriptively statistics | | |
| | following st | andard statistical and e | pidemiological methods. |
| | Approximately 240 patients are expected to be enrolled in the study in a | | |
| | consecutive manner between February 2019 and February 2022 from the | | |
| | participating sites according to the feasibility procedure of the sites. The | | |
| | number of recruited patients as well as the duration of the study is not | | |
| | defined by a formal sample size and power calculation, but is based | | |
| | mainly on the availability of eligible IPF patients as well as patient | | |
| | population in t | he selected sites. | |
| | <u> </u> | | |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingell | heim | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | | Trends in Quality of Life in I<br>th Nintedanib | Patients with IPF Under |
| Study size | Next table des | cribes expected 95% confider | nce limits and precision of the |
| (cont'd): | estimate of me | ean change from baseline of S | GRQ Total Score at week 52, |
| | according to different assumption of mean change from baseline and | | |
| | standard devia | tion (SD). | |
| | Because SD is unknown at the planning stage, it needs to be assumed | | |
| | based on the | previous trials. In INPULSIS | S trials, the sample standard |
| | deviation of the | ne change from baseline in S | GRQ total score at Week 52 |
| | was about 16. | In the real-world setting, the | he more diverse patients are |
| | expected comp | pared to patients in INPULSIS | S trials. These calculations are |
| | based on a total | al number of 200 evaluable st | tudy participants. Taking into |
| | consideration | a withdrawal rate of 17-20% | , the number of patients that |
| | will be enrolled is 240. | | |
| | Therefore, we assume that SD ranging from 16 to 22, as per the table | | |
| | below (95% confidence limits and precision of the estimate of mean | | |
| | change from baseline of SGRQ Total Score at week 52, according to | | |
| | different assu | imption of mean change f | from baseline and standard |
| | deviation): | | |

| Name of compan | ıy: | | | | | |
|---|---|---|---|---|---|---|
| Boehringer Ingell | neim | | | | | |
| Name of finished medicinal | | | | | | |
| product: | | | | | | |
| OFEV | | | | | | |
| Name of active in | ngredient: | | | | | |
| ATC code: L01X | E31 | | | | | |
| Nintedanib | | | | | | |
| Protocol date: | Study | Version/Rev | vision: 3.0 | | Version/Rev | vision date: |
| 11 Sep 2018 | number: | | | | 11 Feb 2021 | |
| | 1199-0355 | | | | | |
| Title of study: | Investigating | Trends in Qua | ality of Lif | fe in Patio | ents with IPF | Under |
| | Treatment wit | th Nintedanib | | | | |
| Study size | N | Mean dif | Sd | 9: | 5% CI | ω |
| (cont'd): | 200 | 2 | 16 | -0.2 | 4.2 | 4.4 |
| | 200 | 2 | 18 | -0.5 | 4.5 | 5.0 |
| | 200 | 2 | 20 | -0.8 | 4.8 | 5.5 |
| | 200 | 2 | 22 | -1.0 | 5.0 | 6.1 |
| | 200 | 3 | 16 | 0.8 | 5.2 | 4.4 |
| | 200 | 3 | 18 | 0.5 | 5.5 | 5.0 |
| | 200 | 3 | 20 | 0.2 | 5.8 | 5.5 |
| | 200 | 3 | 22 | 0.0 | 6.0 | 6.1 |
| | 200 | 4 | 16 | 1.8 | 6.2 | 4.4 |
| | 200 | 4 | 18 | 1.5 | 6.5 | 5.0 |
| | 200 | 4 | 20 | 1.2 | 6.8 | 5.5 |
| | 200 | 4 | 22 | 1.0 | 7.0 | 6.1 |
| | 200 | 5 | 16 | 2.8 | 7.2 | 4.4 |
| | 200 | 5 | 18 | 2.5 | 7.5 | 5.0 |
| | 200 | 5 | 20 | 2.2 | 7.8 | 5.5 |
| | 200 | 5 | 22 | 2.0 | 8.0 | 6.1 |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingel | heim | | |
| Name of finished medicinal | | | |
| product: | | | |
| OFEV | | | |
| Name of active i | ngredient: | | - |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | tients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Data analysis: | Continuous v | rariables will be listed as media | n with interquartile and/or |
| | other percent | iles and as mean value with star | ndard deviation (SD), along |
| | with minimus | m and maximum values and 95 | 5% confidence intervals (if |
| | needed). Cate | egorical values will be summaris | sed as absolute and relative |
| | frequencies. | | |
| | Analysis of P | Primary Outcome | |
| | Summary star | tistics based on observed data v | will be used to describe the |
| | mean SGRQ | scores at each visit and the mea | an change of SGRQ scores |
| | from baseline to each study visit until 12 months. | | |
| | Change from baseline of SGRQ scores will be statistically investigated | | |
| | by mixed mod | dels for repeated measures assur | ning that missing values are |
| | missing at ran | ndom. Baseline is defined as th | e time of the enrolment of |
| | patients in the | e study. | |

| Name of compar | ny: | | |
|---|---|---|---|
| Boehringer Ingell | neim | | |
| Name of finished medicinal | | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | number: | | 11 Feb 2021 |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment wi | th Nintedanib | |
| Data analysis | Analysis of s | econdary outcomes | |
| (cont'd): | Mean change | e from baseline during the 52 | weeks follow up period |
| | (3,6,9,12 mor | nths) for the following endpoints | <b>:</b> : |
| | • burde | n of cough as measured via Coug | gh - Visual Analogue Scale |
| | (Coug | h - VAS) and | |
| | anxiety as me | easured by GAD-7 score, will for | ollow the same analysis as |
| | the primary o | utcome. | |
| | Baseline is de | efined as the time of the enrollme | ent of patients in the study. |
| | Adherence to | nintedanib will be accessed vi- | a frequency tables of each |
| | SMAQ item i | n each follow up visit. | |
| | The number and percentage of patients that use LTOT during the 52 | | |
| | weeks follow up period will also be displayed. The distribution of | | |
| | patients with respect to dyspnoea based on the mMRC score at every | | |
| | study time-po | study time-point, will be presented in frequency tables (N, %). | |

| Name of compar | ıy: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished | l medicinal | | |
| product: | | | |
| OFEV | | | |
| Name of active in | ngredient: | | |
| ATC code: L01X | E31 | | |
| Nintedanib | | | |
| 11 Sep 2018 | <b>number:</b> 11 Feb 2021 | | |
| | 1199-0355 | | |
| Title of study: | Investigating | Trends in Quality of Life in Pat | ients with IPF Under |
| | Treatment with Nintedanib | | |
| Data analysis | Safety Analy | rsis | |
| (cont'd): | All adverse e | vents recorded during the trial w | vill be presented in listings. |
| | AEs will be c | oded based on the MedDRA ter | minology. |
| Milestones: | Study timelin | es depend upon approval of the | final protocol |
| | - feasibil | ity assessment: Sep 2018 | |
| | - IRB/IEC approval: Nov 2018 | | |
| | - start of data collection: Feb 2019 | | |
| | - end of data collection: Mar 2023 | | |
| | - final results: Q3 2023 | | |
| | | udy report: Dec 2023 | |

# 5. AMENDMENTS AND UPDATES

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 1 | 02 June 2020 | 4. ABSTRACT | This is a National, multi-center, non-interventional, prospective cohort study aiming to enroll 240 IPF patients receiving treatment with nintedanib in a consecutive manner from 10-12 reference centers across Greece, representative of the entire Greek population. Recruitment will last for 24 months and patients will be followed over a period of 52 weeks. A baseline visit and 4 follow up visits will be performed during the follow-up period according to clinical practice. | Recruitment period has been extended to 24 months and sample size has been increased to 240 patients, in order for the statistical power and validity of the study's results to get strengthened. |

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 2 | 02 June 2020 | 4. ABSTRACT | mMRC is a modified medical research council dyspnoea scale that uses same descriptors as the original MRC scale. The descriptors of the mMRC scale are numbered 1-5 and are used to estimate the patient's perception of breathlessness. The specific scale has been validated as a measurement of disease severity in IPF patients. | The mMRC description was corrected to reflect its constitution of five descriptors instead of 6. |
| 3 | 02 June 2020 | 4. ABSTRACT | _ | Clarification to Inclusion criterion no 3, on treatment initiation, was added. |

| Number | Date | Section of study protocol | Amendment or update | | Reason |
|---|---|---|---|---|---|
| 4 | 02 June 2020 | 3.<br>RESPONSIBLE<br>PARTIES | Trial Sponsor | BI Greece new address was added. | |
| 5 | 02 June 2020 | 6.MILESTONES | Milestone | Planned Date | Update of the main milestones dates, so that the actual timelines |
| | | | IRB/IEC approval | 14 NOV 2018 | and actual plan to be reflected |
| | | | Start of data collection | 28 FEB 2019 | accurately, based on the visit schedule of the protocol and taking |
| | | | End of data collection | 27 MAR 2022 | into consideration that the first investigational site was activated |
| | | | Final report of study results: | DEC 2022 | on 28 Feb 2019 and the data collection initiated on 28 Feb 2019. |

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 6 | 02 June 2020 | 7.6.1 Rationale for questionnaires used | mMRC is a modified medical research council dyspnoea scale that uses same descriptors as the original MRC scale. The descriptors of the mMRC scale are numbered 1-5 and are used to estimate the patient's perception of breathlessness. The specific scale has been validated as a measurement of disease severity in IPF patients. | The mMRC description was corrected to reflect its constitution of five descriptors instead of 6. |
| 7 | 02 June 2020 | 9.1 STUDY<br>DESIGN | This is a National, multi-center, non-interventional, prospective cohort study aiming to enroll 240 IPF patients receiving treatment with nintedanib in a consecutive manner from 10-12 reference centers across Greece, representative of the entire Greek population. Recruitment will last for 24 months and patients will be followed over a period of 52 weeks. | Recruitment period has been extended to 24 months and sample size has been increased to 240 patients, in order for the statistical power and validity of the study's results to get strengthened. |

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 8 | 02 June 2020 | 9.2.2 Study population | Inclusion Criterion no 3 was updated to: Treatment naïve patients with an initial IPF diagnosis no more than 3 months prior to enrolment according to 2011 ATS/ERS/JRS/ALAT guidelines who are initiating treatment with Nintedanib (as monotherapy for IPF) the latest on the enrollment day or have initiated treatment with Nintedanib (as monotherapy for IPF) within the past 7 days prior to enrolment. | Clarification to Inclusion criterion no 3, on treatment initiation was added. |
| 9 | 02 June 2020 | 9.2.3 STUDY<br>VISITS | The study is scheduled to run for 3 years in total, i.e. 2 years of recruitment and 1 year of follow-up. | Recruitment period extended to 2 years in total and total study duration to 3 years e. g 2 tears recruitment and 1 year of follow up |
| 10 | 02 June 2020 | 9.3.3 Covariates | Long Term Oxygen Therapy: It will be recorded whether the patient is on LTOT or not. | Type and duration of Long-term Oxygen supplementation therapy were deleted, as not required. |

| Number | Date | Section of study protocol | Amendment or update | | | | | Reason | |
|---|---|---|---|---|---|---|---|---|---|
| 11 | 02 June 2020 | Table 1 List of variables to be documented at scheduled visits | Final Visit (12 months follow up ± 1 month or after study discontinuation visit) | | | | | Final Visit definition was updated in Table 1 & Table 2 to better describe study discontinuation visit. | |
| 12 | 02 June 2020 | Table 2 Study<br>Flowchart | Final Visit (12 months follow up $\pm$ 1 month or after study discontinuation visit) | | | | Final Visit definition was updated in Table 1 & Table 2 to better describe study discontinuation visit. | | |
| 13 | 02 June 2020 | 9.5 STUDY<br>SIZE<br>Table 1. 95% | N | Mean<br>dif | Sd | 95% CI Ω | | Ω | Inclusion of the newly calculated confidence intervals, based on the new sample size into a revised Table |
| | | confidence limits | 200 | 2 | 16 | -0.2 | 4.2 | 4.4 | 3. |
| | | and precision of | 200 | 2 | 18 | -0.5 | 4.5 | 5.0 | |
| | | the estimate of mean change from | 200 | 2 | 20 | -0.8 | 4.8 | 5.5 | |
| | | baseline of SGRQ | 200 | 2 | 22 | -1.0 | 5.0 | 6.1 | |
| | | Total Score at | 200 | 3 | 16 | 0.8 | 5.2 | 4.4 | |
| | | week 52, according to different | 200 | 3 | 18 | 0.5 | 5.5 | 5.0 | |
| | | assumption of | 200 | 3 | 20 | 0.2 | 5.8 | 5.5 | |
| | mean change from baseline and standard deviation. | | | | | | | | |
| Number | Date | Section of study protocol | Amendment or update | | | | | | Reason |
|---|---|---|---|---|---|---|---|---|---|
| 13 (cont'd) | 02 June 2020 | 9.6 STUDY SIZE Table 1. 95% | N | Mean<br>dif | Sd | 95% | 6 CI | Ω | Inclusion of the newly calculated confidence intervals, based on the new sample size into a revised Table |
| | | confidence limits and precision of | 200 | 3 | 22 | -0.0 | 6.0 | 6.1 | 3. |
| | | the estimate of | 200 | 4 | 16 | 1.8 | 6.2 | 4.4 | |
| | | mean change from | 200 | 4 | 18 | 1.5 | 6.5 | 5.0 | |
| | | baseline of SGRQ Total Score at | 200 | 4 | 20 | 1.2 | 6.8 | 5.5 | |
| | | week 52, according | 200 | 4 | 22 | 1.0 | 7.0 | 6.1 | |
| | | to different | 200 | 5 | 16 | 2.8 | 7.2 | 4.4 | |
| | | assumption of mean change from | 200 | 5 | 18 | 2.5 | 7.5 | 5.0 | |
| | | baseline and | 200 | 5 | 20 | 2.2 | 7.8 | 5.5 | |
| | | standard deviation. | 200 | 5 | 22 | 2.0 | 8.0 | 6.1 | |
| | | | | 1 | 1 | <u> </u> | 1 | | |

| Number | Date | Section of study protocol | Amendment or update | | Reason |
|---|---|---|---|---|---|
| 14 | 02 June 2020 | ANNEX 3:<br>ADDITIONAL<br>INFORMATION | mMRC descriptor was correct was for breath after walk after a few minutes on the left of the form of the left of the few minutes on the left of the few minutes of the | king about 100 <b>yards</b> or<br>evel" instead of<br>king about 100 <b>meters</b> or | Corrected mMRC U.S version added to include at the descriptor yards instead of meters: "I stop for breath after walking about 100 yards or after a few minutes on the level" |
| 15 | 11 Feb 2021 | 6. MILESTONES | Milestone | Planned Date | Update of the main milestones |
| | | | IRB/IEC approval | 14 NOV 2018 | dates, to reflect the extended timelines. |
| | | | Start of data collection | 28 FEB 2019 | |
| | | | End of data collection | 27 MAR 2023 | |
| | | | Final report of study results: | DEC 2023 | |

# 6. MILESTONES

| Milestone | Planned Date |
|--------------------------------|--------------|
| IRB/IEC approval | 14 NOV 2018 |
| Start of data collection | 28 FEB 2019 |
| End of data collection | 27 MAR 2023 |
| Final report of study results: | DEC 2023 |

## 7. RATIONALE AND BACKGROUND

## 7.1 **DEFINITION**

Idiopathic pulmonary fibrosis (IPF) is defined as a specific form of chronic, progressive fibrosing interstitial pneumonia of unknown cause, occurring primarily in older adults, limited to the lungs (2). It is characterized by progressive worsening of dyspnea and lung function and is associated with a poor prognosis. As stated in an international consensus statement jointly issued by ATS/ERS, JRS and ALAT, IPF is a distinct clinical entity associated with the histologic and/or radiologic appearance of usual interstitial pneumonia (UIP) (2). The definition of IPF requires the exclusion of other forms of interstitial pneumonia including other idiopathic interstitial pneumonias (IIP) and interstitial lung disease (ILD) associated with environmental exposure, medication, or systemic disease (2).

IPF predominantly presents in older individuals (cases in persons aged less than 50 years are rare), with a preponderance in men and previous or current smokers. Patients present with unexplained chronic exertional dyspnea, and commonly with cough, bibasilar inspiratory crackles, and finger clubbing.

# 7.2 INCIDENCE AND PREVALENCE

Overall, epidemiological data on the incidence and prevalence of IPF are limited, as stated in the consensus statement issued by ATS/ERS/JRS/ALAT (2). IPF prevalence varies widely between 1.25 and 63 cases per 100,000 of population in several epidemiological studies (1, 3, 9-12). Incidence of IPF is also variable. A systematic review reported an incidence range of 2.8-9.3 per 100,000 population per year in Europe and North America (1). In this analysis, it was noted that there was an increase in IPF incidence over time according to most studies, but mortality appears to plateau and even decline in USA and Denmark (13, 14). Regarding Greece, Karakatsani et al conducted a multicenter survey in 2009, using an one page questionnaire, in order to evaluate the incidence and prevalence of Interstitial Lung Diseases in Greece (10). Centers covering about 60% of Greek population were analyzed. A total of 967 cases of ILDs were registered. The most frequent disease was sarcoidosis (34.1%), followed in decreasing order by IPF (19.5%). The annual incidence of IPF was estimated to be 0.93 cases per 100,000, whereas prevalence was estimated to be 3.38 cases per 100,000. Since then though, the

diagnostic criteria, the international guidelines, the standard medical care and the composition of the population have changed and possibly these data do not reflect the current population of IPF patients (2, 5, 15).

#### 7.3 DIAGNOSIS

According to the consensus statement jointly issued by ATS/ERS/JRS/ALAT in 2011, the diagnosis of IPF requires the following (2):

- Exclusion of other known causes of ILD (e.g., domestic and occupational environmental exposures, connective tissue disease, and drug toxicity).
- The presence of a UIP pattern on HRCT in patients not subjected to surgical lung biopsy.
- Specific combinations of HRCT and surgical lung biopsy pattern in patients subjected to surgical lung biopsy.

#### 7.4 NATURAL COURSE

Data on the natural course of IPF are from retrospective and a few prospective studies, including the placebo arms of clinical trials (limited to short observation periods and by in-/exclusion criteria). The previously reported median survival time of 2-3 years from the time of diagnosis could be an underestimate, at least when accounting for patients with preserved lung function. Notably, the natural course is unpredictable for a given patient at the time of diagnosis, while the majority of patients experience steady worsening (slow progression), other remain stable, or have rapid progression of disease (9, 10). Acute respiratory worsening either due to secondary complications (e.g. pneumonia, pulmonary embolism, pneumothorax or cardiac failure) or due to unknown reasons (in this case the term acute exacerbation is used) are suggested to occur in about 5-10% annually (2, 16, 17). A recent retrospective review of 461 patients with IPF has found that the 1- and 3-year incidences of acute exacerbations were 14.2% and 20.7%, respectively (10).

## 7.5 THERAPY

Until recently, there was no effective pharmacological treatment for IPF, other than lung transplantation that was considered the only survival improving intervention. Since 2011, two novel agents, pirfenidone and nintedanib, have been approved by both EMA and FDA for patients with IPF, on the basis of phase III randomized clinical trials (RCTs) showing that these agents reduce the decline of lung function in comparison to placebo (18-21).

Nintedanib is a multi-target tyrosine kinase inhibitor with activity against vascular endothelial growth factor (VEGF), fibroblast growth factor (FGF), and platelet-derived growth factor (PDGF) receptors, that are implicated in the pathogenesis of IPF (22, 23). Three RCTs – one phase 2 study (TOMORROW) and two replicate phase 3 studies (INPULSIS-1 and INPULSIS-2) – have been conducted to evaluate efficacy of nintedanib in IPF (20, 21). The two phase 3 trials met their primary endpoint showing that nintedanib at a dose of 150mg twice daily reduced statistically significant the adjusted annual rate of decline in FVC (21). Furthermore, pooled analysis of all three RCTs conducted with nintedanib in IPF showed a trend for reduced mortality and statistically significant reduction in the number of acute exacerbations among IPF patients treated with nintedanib (20, 21).

Both drugs have also received conditional recommendation for use according to the latest ATS/ERS/JRS/ALAT clinical practice guidelines for IPF (15).

## 7.6 RATIONALE FOR THE PRESENT STUDY

Due to the rarity of IPF, there are very limited data regarding the patients' population, the natural course of the disease and the medical treatment these patients receive, as highlighted by the call for action towards a worldwide IPF registry (5). Especially for the Greek population, very few data are available regarding the use of nintedanib in cohorts of patients with IPF either pre-treated or treatment-naïve, also in terms of Patients Reported Outcomes (PRO) (6). The recently launched observational study INDULGE-IPF (NCT03074149) will provide

essential data regarding the natural course of IPF and the treatment of the disease – including the use of nintedanib – in the Greek population.

In a chronic disease like IPF, the goal of pharmacological treatments should not be only survival prolongation, but also delay in the progression of the disease and on the clinical deterioration of patients, i.e. delay in worsening of symptoms and quality of life. In IPF there is a paucity of well validated PRO measures. In the pooled analysis of nintedanib randomized trials in IPF, the use of SGRQ questionnaire as a measurement of health related quality of life provided evidence for a modest effect of nintedanib on the delay of clinical deterioration of patients (4, 7). In addition a German IPF registry (INSIGHTS-IPF) has recently published results for patient reported outcomes (PROs) in enrolled patients, showing IPF patients under real-life conditions have lower HRQoL compared to those in clinical studies (8). In the Greek population though, analogous results regarding the effect of nintedanib on SGRQ as well as other PRO measures are lacking.

In pharmacological treatments, efficacy is of outmost importance. In chronic diseases like IPF, the approval of a new effective treatment may lead to long-term exposure to the drug. This is beneficial in terms of disease outcomes for the patients but may also be accompanied by adverse events associated with the prolonged use of the treatment. IPF is a progressive disease and current treatments have shown to slow disease progression. In addition, randomized clinical trials with nintedanib have shown that the drug did not adversely affect the quality of life of the patients at least as this was evaluated by the SGRQ questionnaire. However, detailed description of the several parameters related with the quality of life of IPF patients under treatment with nintedanib may provide further insight for the optimal use of the drug and the appropriate management of the patients. Furthermore, such data could provide clinicians with valuable information related to the anticipated evolution of the quality of life of IPF patients under nintedanib treatment.

# 7.6.1 Rationale for questionnaires used

In this study, PROs will be used in a cohort of newly diagnosed IPF patients that have recently started treatment with nintedanib in order to provide relevant information regarding IPF-related symptoms and their impact on several aspects of everyday life activities including

psychological consequences. Periodical completion of PROs will allow to record in this cohort of patients' evolution of IPF symptoms and their effects on HRQoL. Finally, adherence to treatment will be recorded. Patients will be reporting on very specific symptoms (e.g., cough, dyspnoea) and their functional impact, which are concepts proximal to patients' experience with the disease and treatment. Although an assessor bias cannot be disregarded in an openlabel setting, it is unlikely that this bias would be of such magnitude as to invalidate the data collected through PROs.

Instruments implemented in the study - namely the St George's Respiratory Questionnaire (SGRQ) (24), the modified Medical Research Council scale (mMRC) (25), the Cough - Visual Analogue Scale (Cough - VAS), the Simplified Medication Adherence Questionnaire (SMAQ) (26) and Generalized Anxiety Disorder 7-item scale (GAD-7) (27) - have been selected on the basis of their content validity and performance and to minimize patients' completion burden.

More specifically SGRQ is a self-administered, 50-item questionnaire assessing three domains: symptoms, activity and impact. The symptoms domain addresses the frequency and severity of respiratory symptoms; the activity domain assesses activities that cause or are limited by breathlessness and the impact domain taps a range of aspects concerned with social functioning and the psychological impact of the disease. SGRQ was initially developed for use in patients with COPD or asthma (24), but has also been used for IPF patients (4, 28). The total SGRQ score and the score for each domain range from 0 to 100, with higher scores indicating worse health-related quality of life. A minimally important difference in the score has not been established for patients with idiopathic pulmonary fibrosis; in patients with chronic obstructive pulmonary disease, this difference is 4 points.

Analogously, mMRC is a modified medical research council dyspnoea scale that uses same descriptors as the original MRC scale. The descriptors of the mMRC scale are numbered 1-5 and are used to estimate the patient's perception of breathlessness. The specific scale has been validated as a measurement of disease severity in IPF patients(29).

Cough - VAS has been used as an easy and fast method to assess intensity of IPF related cough and is a recommended instrument for IPF patients (30).

SMAQ is a six-item questionnaire that estimates in a qualitative and semi-quantitative manner the adherence of patients to treatment. SMAQ has already been validated for several medical and non-medical interventions (26).

Finally, GAD-7 is a 7-item instrument validated for anxiety evaluation that could be used in outpatient setting.

# 8. RESEARCH QUESTION AND OBJECTIVES

The aim of this non-interventional-study based on newly collected data is to collect data on various important PROs in patients with IPF that could provide useful insights about HRQoL over 52 weeks in patients treated with nintedanib in the real world setting in Greece.

# Primary objective:

• To evaluate changes from baseline of HRQoL for IPF patients treated in current clinical practice in Greece with nintedanib at time-points of 3, 6, 9 and 12 months over a 52-weeks period, via SGRQ (For a sample of the English version please refer to <u>ANNEX 3: SGRQ</u>).

# Secondary objectives are:

- To assess changes, from baseline, in dyspnoea and cough in IPF patients treated with nintedanib in current clinical practice in Greece at time-points of 3, 6, 9 and 12 months over a 52 weeks period, via specific questionnaires, such mMRC score (For sample of the English version please refer to <u>ANNEX 3: mMRC</u>) and Cough Visual Analogue Scale (Cough VAS) respectively (For sample of the English version please refer to <u>ANNEX 3: Cough VAS</u>).
- To estimate the adherence to nintedanib treatment in current clinical practice at time-points of 3, 6, 9 and 12 months over a 52 weeks period via SMAQ Questionnaire (adapted for the treatment of idiopathic pulmonary fibrosis (IPF)) (For a sample of the English version please refer to ANNEX 3: SMAQ).
- To measure anxiety in IPF patients treated with nintedanib in current clinical practice in Greece at time-points of baseline, 3, 6, 9 and 12 months over a 52 weeks period via GAD-7 Questionnaire (For a sample of the English version please refer to ANNEX 3: GAD-7).
- To estimate the use of Long Term Oxygen Treatment (LTOT) among IPF patients under treatment with nintedanib in current clinical practice in Greece at time-points of baseline, 3, 6, 9 and 12 months over a 52 weeks period.

## 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is a National, multi-center, non-interventional, prospective cohort study aiming to enroll 240 IPF patients receiving treatment with nintedanib in a consecutive manner from 10-12 reference centers across Greece, representative of the entire Greek population. Recruitment will last for 36 months and patients will be followed over a period of 52 weeks. Only consecutive patients with newly diagnosed IPF patients (initial IPF diagnosis no more than 3 months prior to enrolment) according to 2011 ATS/ERS/JRS/ALAT guidelines who are initiating treatment with nintedanib will be enrolled to restrict selection bias. A baseline visit and estimated 4 follow up visits will be performed during the follow-up period according to clinical practice. In the context of this study, participating physicians shall follow each enrolled patient for a planned observation period of 12 months, starting from the date of baseline visit and ending at the earliest of treatment discontinuation, withdrawal of consent, physician's decision to withdraw the patient, 12-month observation period completion, death or any other discontinuation criterion is met.

Patients that permanently discontinue nintedanib treatment for any reason (e.g. due to AE, consent withdrawal, lost to Follow-up) prior to the follow up period completion, will no longer be followed-up for the study and the visit that nintedanib discontinuation is recorded will be considered as their end of study visit.

# 9.2 SETTING

## 9.2.1 Study sites

This is a National multicenter study that will enroll patients in 10-12 sites, academic hospitals and reference centers. All included sites are reference centers for IPF. Furthermore, sites both in Athens and rest of Greece are included in the study so as patients enrolled will constitute a representative population of IPF patients in Greece.

# 9.2.2 Study population

Newly diagnosed IPF patients initiating treatment with nintedanib according to their physician's clinical decision will be enrolled in this study. In details, patients will be eligible to enroll in the study if the fulfil all the inclusion criteria and none of the exclusion criteria:

#### **Inclusion criteria**

- Patients  $\geq$ 40 years of age.
- Patients that have signed Informed Consent Form.
- Treatment naive patients with an initial IPF diagnosis no more than 3 months prior to enrolment according to 2011 ATS/ERS/JRS/ALAT guidelines who are initiating treatment with nintedanib (as monotherapy for IPF), the latest on the enrollment day or have initiated treatment with nintedanib (as monotherapy for IPF) within the past 7 days prior to enrolment.
- Patients for whom the decision to prescribe therapy with nintedanib according to the
  locally approved product's Summary of Product Characteristics (SmPC) has already been
  taken prior to their enrolment in the study and is clearly separated from the physician's
  decision to include the patient in the current study.
- Patients that are able to read, understand and complete the study specific questionnaires.

#### **Exclusion criteria**

- Treatment with nintedanib for more than 7 days prior to study enrolment.
- Patients receiving a combination therapy of nintedanib & pirfenidone for IPF.
- Patients that meet any of the contraindications to the administration of the study drug nintedanib according to the approved SmPC.
- Prior treatment with pirfenidone or other treatment for IPF.
- Participation in an interventional study.
- Patients currently receive treatment with any investigational drug/device/intervention or have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) before the initiation of therapy with nintedanib.

According to study design, enrolled patients will constitute a representative population of newly diagnosed IPF patients in Greece. Recruitment will last for 36 months and patients will be followed over a period of 52 weeks post enrollment. A baseline visit and estimated 4 follow up visits will be performed during the follow-up period according to clinical practice. Patients will be included in a consecutive manner at each site between February 2019 and February 2022 in order to avoid selection bias.

A subject screening log should be kept at the site, recording basic information (e.g. initials, gender, date of birth, reason for not enrolling the patient etc.) on all patients who were invited to participate in the study, with the information on the eligibility (or reasons for non-eligibility) and date of signed informed consent. In the case of refusal, reasons for refusal should be given. In addition, a log of all patients included into the study (i.e. having given informed consent) will be maintained in the study file at the study site.

## 9.2.3 Study visits

The study is scheduled to run for 4 years in total, i.e. 3 years of recruitment and 1 year of follow-up. During the follow up period, data will be collected on 4 standard clinical visits which usually are scheduled around: 3-months ( $\pm$  1 month), 6-months ( $\pm$  1 month), 9-months ( $\pm$  1 month), 12-months ( $\pm$  1 month) until the end of participation in the study. Patients that permanently discontinue nintedanib treatment for any reason (e.g. due to AE, consent withdrawal, lost to Follow-up) prior to the follow up period completion, will no longer be followed-up for the study and the visit that nintedanib discontinuation is recorded will be considered as their end of study visit.

#### 9.2.4 Patient discontinuation

Patients will be followed up for a 52-weeks follow-up period according to clinical practice and will be considered that completed the study upon completion of the last FU data collection at week 52. Patients that withdraw from the study prior to the follow up period completion, for any reason (consent withdrawal, lost to follow up) will no longer be followed-up for the study and the visit that discontinuation is recorded will be considered as their final, end of study visit.

**BI Study Number 1199-0355** 

Proprietary confidential information © 2021BoehringerIngelheim International GmbH or one or more of its affiliated companies

In case of patient's permanently treatment discontinuation for any reason (e.g. due to AE, physician's decision), patients will be considered as prematurely/early discontinued and will not be further followed up in the scope of the study. The visit that discontinuation is recorded will be considered as their final, end of study visit.

Patients that temporarily interrupt treatment with nintedanib, up to 28 days, will continue follow up activities according to the study plan and will not be discontinued from the study. In case of dose reduction during the course of the study and re-start, patients will continue their participation and information on treatment administration will continue to be captured (dose reduction, treatment re-start and dose).

Patients reserve the right to discontinue their participation in the study at any time during its conduct and for any reason, without having to justify their decision and with no impact on their future medical care and therapy.

Consent withdrawal means that a patient does not want or is unable to further continue participating in the study.

The reasons for patient's discontinuation may include the following:

- patient's withdrawal of informed consent;
- discontinuation of study treatment (nintedanib) due to any reason;
- the patient meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation;
- enrollment or planned participation in any clinical trial, at any time during the study observation period, in which the patient has been or will be exposed to an investigational product (pharmaceutical agent or device) or intervention;
- investigator's/physician's decision;
- significant protocol deviation/violation.

Patients, who withdraw from the study, should be asked about the reason(s) for discontinuation and the occurrence of any adverse events, and, if applicable, they shall be examined and evaluated by the investigator as per the procedures defined in the Final / Discontinuation Visit.

Furthermore, investigators will have the right to withdraw any patient from the study, if according to their clinical judgment this decision is considered to be in the patient's best interest.

If a patient withdraws or is removed from the study for any reason, the reason for and date of the discontinuation as well as the date of the last dose of study medication should be recorded in the appropriate section of the electronic Case Report Form (eCRF).

## 9.2.5 Study discontinuation

Boehringer Ingelheim reserves the right to discontinue the study overall or at a particular study site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular study site
- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the study, or any other administrative reasons.
- 3. Violation of Good Clinical Practice (GCP) (as applicable), Good Pharmacoepidemiology Practice (GPP), the study protocol, or the contract by a study site or investigator, disturbing the appropriate conduct of the study

The investigator / the study site will be reimbursed for reasonable expenses incurred in case of study termination (except in case of the third reason).

#### 9.3 VARIABLES

## 9.3.1 Exposures

All patients included in the study will receive nintedanib based on the clinical decision of their treating physician. Normally nintedanib standard dose is 150mg twice daily, as per the SmPC. It is possible to reduce the dose of nintedanib to 100mg twice daily in case of intolerance.

Patients will be followed up until end of study period (in case they receive treatment with nintedanib for a 52-weeks follow-up period according to clinical practice) or until discontinuation. In case of dose reduction this information will be captured and patients will continue to be followed-up in the study.

# 9.3.2 Endpoints

# 9.3.2.1 Primary endpoint

The primary endpoint of the study is:

• The mean change from baseline in HRQoL (with reference to SGRQ score, both total score and score in each of the SGRQ domains) of patients under treatment with nintedanib, as assessed by the changes in SGRQ score at time-points of 3, 6, 9 and 12 months over the 52 weeks follow-up period.

# 9.3.2.2 Secondary endpoints

The secondary endpoints of the study are:

- The mean change from baseline to 3, 6, 9 and 12 months follow up period of dyspnoea burden, as measured via changes in the mMRC score
- The mean change from baseline to 3, 6, 9 and 12 months follow up period of cough burden, as measured via changes in the Cough Visual Analogue Scale (Cough VAS).
- Percentage of adhered patients to nintedanib treatment at time-points of 3, 6, 9 and 12 months over the 52 weeks follow up period, as measured via SMAQ questionnaire (adapted for the treatment of idiopathic pulmonary fibrosis (IPF).
- The mean change from baseline to 3, 6, 9 and 12 months follow up period of anxiety in patients treated with nintedanib, as measured via GAD-7 questionnaire.
- Percentage of patients that use LTOT at time-points of 3, 6, 9 and 12 months over the 52 weeks follow up period.



#### 9.3.3 Covariates

Due to the non - interventional nature and design of this study, it does not require strict timeline visit schedule. Patients will receive treatment with nintedanib according to standard clinical practice with regards to approximate visit frequencies described above, type of performed assessments and according to local prescription requirements.

Following identification of a potential patient, the investigator will follow the below listed procedures:

- 1. Review of individual patient's medical history, to confirm that the inclusion/exclusion criteria are met.
- 2. Explanation of the study objectives to the patient and receipt of signed and dated informed consent, after providing the patient with sufficient time to read carefully and understand the information sheet.
- 3. Data collection from the medical records of eligible for enrollment patients, as required by eCRF, and eCRF completion.

Please refer to <u>Section 11.2</u> for details regarding Adverse Event and Serious Adverse Event Collection and Reporting.

A tabulated schedule of assessments that provide information regarding the recommended timeline of data collection and represents the standard clinical care of IPF treated patients is listed below in <u>Table 1</u>. The exact definitions of the variables are the following:

- Basic (Socio-) demographic data. Age (date of birth), gender (sex), race
- Anthropometric characteristics. Height and weight of the patients will be recorded

- Physical and vital signs examination. Blood pressure (sitting systolic and diastolic arterial pressure), and heart rate will be recorded
- IPF risk factors. These include smoking habit (past or current smoker, non-smoker or unknown) and number of pack-years, environmental and occupational exposure; alcohol and substance abuse, exposure to drugs associated with pulmonary fibrosis, exposure to viral infection possibly related to IPF, gastro-esophageal reflux, genetic factors (family history), or others.
- Co-morbidities and concomitant treatments (medication category/class).
- Date and method of IPF diagnosis. Dates and results of High Resolution Chest CT (HRCT), surgical lung biopsy and bronchoalveolar lavage will be recorded if already performed
- IPF symptoms. Presence of dyspnea, cough, fatigue, dizziness, chest pain and anxiety as reported by the patient will be recorded.
- Nintedanib treatment. Start date and stop date, dates of treatment interruption, dose reductions and dose re-escalations will be recorded
- Assessment of lung function and exercise capacity. Data recording FVC, DLCO and 6-minutes walking test will be recorded at baseline if already performed.
- Questionnaires. The following questionnaires will be completed by the enrolled patients prior to any clinical assessment at each visit of the study (baseline, follow-up visits and final visit): SGRQ, mMRC Score, Cough VAS and GAD-7. SMAQ questionnaire (adapted for the treatment of idiopathic pulmonary fibrosis (IPF) will be completed by the enrolled patients prior to any clinical assessment at each follow-up visit of the study.
- Long Term Oxygen Therapy, . It will be recorded whether the patient is on LTOT or not.
- Survival status. Patient dead or alive.

Table 1 List of variables to be documented (if available) at scheduled visits

| Variable | Assessment | Follow up 1-3* | Final Visit (12 months follow up ± 1 month or study discontinuation visit) |
|---|---|---|---|
| Eligibility criteria | X | | |
| Baseline information (ass | sessment) | | |
| (Socio-)demographic variables: age (date of birth), gender, race | X | | |
| Anthropometric characteristics: height | X | | |
| Anthropometric characteristics: body weight | X | X | X |
| Physical examination: Blood pressure (sitting systolic and diastolic arterial pressure), heart rate | 11 | Х | X |
| (Possible) IPF risk fa | ectors | | |
| Cigarette smoking incl. pack years (Categorized as never/past/current/unknown. For past/current, specify packs/year and for past, number of years smoking one pack per day); environmental and occupational exposure; alcohol and substance abuse; exposure to drugs associated with pulmonary fibrosis; exposure to viral | X | | |

| oesophageal reflux; genetic factors (family | | | |
|---|---|---|---|
| history); others | | | |
| Co-morbidities | X | | |
| Concomitant medications (changes in concomitant medications in follow ups) | Х | Х | х |
| IPF | | | |
| Baseline information (assessr | ment) on IPF | | |
| First symptoms; date of first diagnosis, dates and results of HRCT, surgical lung biopsy, bronchoalveolar lavage. | Х | | |
| Symptoms | Symptoms | | |
| Dyspnea, cough, fatigue, dizziness, chest pain, anxiety | X | Х | х |
| Functional assessm | ent | | |
| Lung function test (FVC, DLCO) 6-minute walk distance | Х | | |
| Treatment with Nintedanib (start date, stop date, restart date in case of temporary discontinuation and daily dose) | X | Х | Х |
| Long-Term-Oxygen-Therapy (liquid and/or concentrate) | Х | Х | х |
| Questionnaires | | | |
| SGRQ | X | X | х |
| mMRC | X | X | Х |

| Cough - VAS | х | X | Х |
|--------------------------------------|---|---|---|
| GAD-7 | Х | X | Х |
| SMAQ | | X | Х |
| Survival status | | X | Х |
| Reason for treatment discontinuation | | | Х |

For abbreviations, please refer to glossary.

## 9.4 DATA SOURCES

The study will mainly include the recording of new data through a web-based system for data collection. Data will be collected by the study doctors as they occur according to standard clinical practice in the approximate visiting schedule indicated above.

Source (primary) patient data related to their medical and IPF history will be collected by the investigators from the patient's medical files/records and will be documented in the relevant eCRF section.

Data regarding treatment modifications, concomitant treatments, study related routine clinical assessments, and survival status will also be collected. The procedures that should be performed at each study visit are presented as a study flow chart in <u>Table 2</u>.

<sup>\*3-</sup>months ( $\pm$  1 month), 6-months ( $\pm$  1 month), 9-months ( $\pm$  1 month),

<sup>\*\*</sup> Final visit is designated as either the 12 months (± 1 month) follow up visit for all patients that remain on study until that time-point or the visit performed at the time of a patient's discontinuation or withdrawal from the study.

Table 2Study flow chart

| | - ·· | 7774 | | | <b>7.</b> 4 |
|---|---|---|---|---|---|
| | Baseline | FU1 | FU2 | FU3 | Final visit (12 |
| | visit | 3-month | 6-month | 9-month | months follow- |
| | | follow- | follow-up | follow-up | up visit ± 1 |
| | | up visit ± | visit (± 1 | visit (± 1 | month or after |
| | | 1 month) | month) | month) | study |
| | | | | | discontinuation |
| | | | | | visit) |
| Inclusion/exclusion | X | | | | |
| criteria | | | | | |
| ICF signed | X | | | | |
| Sociodemographic | X | | | | |
| variables (age/date of | | | | | |
| birth, gender, race) | | | | | |
| Anthropometric | X | X | X | X | X |
| characteristics (body | | | | | |
| weight) | | | | | |
| Anthropometric | X | | | | |
| characteristics | | | | | |
| (height) | | | | | |
| Physical examination | X | X | X | X | X |
| Blood pressure | X | X | X | X | X |
| (sitting systolic and | | | | | |
| diastolic arterial | | | | | |
| pressure), heart rate | | | | | |
| Completion of | X | X | X | X | X |
| Questionnaires | | | | | |
| (SGRQ, mMRC, | | | | | |

| Cough - VAS, GAD-7) | | | | | |
|---------------------------------------|---|---|---|---|---|
| , | | | | | |
| Completion of | | X | X | X | X |
| SMAQ Questionnaire | | | | | |
| Comorbidities | X | | | | |
| Concomitant | X | X | X | X | X |
| medication | | | | | |
| (medication | | | | | |
| category/class) | | | | | |
| Treatment with | X | X | X | X | X |
| nintedanib | | | | | |
| Clinical evaluation | X | X | X | X | X |
| Survival status | X | X | X | X | X |
| Adverse events | X | X | X | X | X |
| collection and | | | | | |
| recording | | | | | |

## 9.5 STUDY SIZE

This observational study will be analyzed descriptively following standard statistical and epidemiological methods. Approximately 240 patients are expected to be included in the study in a consecutive manner between February 2019 and February 2022 from the participating sites according to the feasibility procedure of the sites. The number of included patients as well as the duration of the study is not defined by a formal sample size and power calculation, but is based mainly on the availability of eligible IPF patients as well as patient population in the selected sites.

<u>Table 3</u> describes expected 95% confidence limits and precision of the estimate of mean change from baseline of SGRQ Total Score at week 52, according to different assumption of mean

change from baseline and standard deviation (SD). Sample size is assumed to be 200 because it is expected that some patients discontinue nintedanib treatment prior to the follow-up period completion.

Because SD is unknown at the planning stage, it needs to be assumed based on the previous trials. In INPULSIS trials, the sample standard deviation of the change from baseline in SGRQ total score at Week 52 was about 16. In the real-world setting, the more diverse patients are expected compared to patients in INPULSIS trials. Therefore, we assume that SD may range from 16 to 22. These calculations are based on a total number of 200 evaluable study participants. Taking into account an approximate dropout rate of 17-20%, a final number of 240 patients will be enrolled in the study.

**Table 3** 95% confidence limits and precision of the estimate of mean change from baseline of SGRQ Total Score at week 52, according to different assumption of mean change from baseline and standard deviation.

| N | Mean dif | Sd | 95% CI | | ω |
|-----|----------|----|--------|-----|-----|
| 200 | 2 | 16 | -0.2 | 4.2 | 4.4 |
| 200 | 2 | 18 | -0.5 | 4.5 | 5.0 |
| 200 | 2 | 20 | -0.8 | 4.8 | 5.5 |
| 200 | 2 | 22 | -1.0 | 5.0 | 6.1 |
| 200 | 3 | 16 | 0.8 | 5.2 | 4.4 |
| 200 | 3 | 18 | 0.5 | 5.5 | 5.0 |
| 200 | 3 | 20 | 0.2 | 5.8 | 5.5 |
| 200 | 3 | 22 | 0.0 | 6.0 | 6.1 |
| 200 | 4 | 16 | 1.8 | 6.2 | 4.4 |
| 200 | 4 | 18 | 1.5 | 6.5 | 5.0 |
| 200 | 4 | 20 | 1.2 | 6.8 | 5.5 |
| 200 | 4 | 22 | 1.0 | 7.0 | 6.1 |
| 200 | 5 | 16 | 2.8 | 7.2 | 4.4 |
| 200 | 5 | 18 | 2.5 | 7.5 | 5.0 |

| 200 | 5 | 20 | 2.2 | 7.8 | 5.5 |
|-----|---|----|-----|-----|-----|
| 200 | 5 | 22 | 2.0 | 8.0 | 6.1 |

## 9.6 DATA MANAGEMENT

This study will include the collection of new data that will be recorded in an existing web-based database in a consecutive manner (electronic case report form, eCRF) as well as transferring already existing data to the system from medical charts. The patients will be identified by subject identification number, site number, and study identification number.

Investigators will enter the data of their patients directly into an internet-based electronic case record form. At data entry, plausibility checks (e.g., range checks, conditional checks, etc.) will be performed. Data will be entered in the eCRF system by the study personnel at the Investigator's site, according to the Investigator Instructions Manual. Data entered in the eCRF system will be automatically saved to a central database and changes tracked to provide an audit trail. When data have been entered, reviewed and edited, the Investigator shall sign the e-CRF electronically as per the agreed project process and data will be locked to prevent further editing.

Query management will be performed through built-in query management functionality that will be incorporated into the eCRF.

Prior to the onset of data management activities, a detailed data management plan (DMP) will be issued describing the procedure to be followed for processing all collected study data in order to ensure they are valid, complete and accurate for statistical analysis. In addition, aiming at ensuring the expected quality of data, a thorough data cleaning session will be applied. When all data have been properly validated and the quality control procedure has been completed, a declaration of database lock will take place so that it can be confirmed that all important actions have been properly performed. In addition, prior to database lock and prior to the initiation of any statistical analysis activities a comprehensive statistical analysis plan (SAP) will be drafted.

The SAP will also include information regarding the statistical software(s) to be used for the analysis of the study data.

#### 9.7 DATA ANALYSIS

## 9.7.1 Main analysis

The objective of this study is neither to confirm nor to reject any predefined hypothesis; therefore, the nature of the statistical analyses will be exploratory and descriptive.

Continuous variables will be listed as median with interquartile and/or other percentiles, and as mean value with standard deviation (SD), along with minimum and maximum values and 95% confidence intervals (if needed). Categorical values will be summarized as in absolute and relative frequencies.

In terms of missing data, any reasonable attempt will be undertaken to ensure completeness of data collection in this study. Imputation of missing values will not be performed. Missing values will be differentiated from negative answers.

## **Analysis of Primary Outcome**

Summary statistics based on observed data will be used to describe the SGRQ scores at each visit and the change of SGRQ scores from baseline to each study visit until week 52.

Evaluation of SGRQ total score and each domain score regarding change from baseline until each study visit, will be performed by mixed models for repeated measures, assuming that missing values are missing at random. Modelling details will be provided in the SAP.

Baseline is defined at time patient is enrolled in the study.

## Analysis of secondary outcomes

Mean change from baseline during the 52 weeks follow up period (3, 6, 9, 12 months) for the following endpoints:

- burden of cough as measured via Cough Visual Analogue Scale (Cough VAS) and
- anxiety as measured by GAD-7 score,

will follow the same analysis as the primary outcome.

Baseline is defined at time patient is enrolled in the study.

Adherence to nintedanib will be accessed via frequency tables (n, %) of each SMAQ item in every follow up visit.

The number and percentage of patients that use LTOT during the 52 weeks follow up period will also be displayed.

The distribution of patients with respect to dyspnoea based on the mMRC score at every study time-point, will be presented in frequency tables (N, %).

# **Safety Analysis**

All adverse events recorded during the trial will be presented in listings. AEs will be coded based on the MedDRA terminology.

# 9.8 QUALITY CONTROL

In order to ensure the quality and integrity of data throughout the course of the study, proper quality control mechanisms and methods will be applied. All procedures will be described in detail in the study specific Data Management Plan (DMP) and Statistical Analysis Plan (SAP).

eCRF files from each participating site will be stored in CD-ROMs after completion of the study and will be distributed to the participating sites.

**BI Study Number 1199-0355** 

Proprietary confidential information © 2021BoehringerIngelheim International GmbH or one or more of its affiliated companies

The investigators will be provided with a folder/file by the authorized representative of the study, in which they will be required to keep and store all study related documents. All study documents will be stored in this file by the Investigator. The contents of this file/folder may be subjected to audit/inspection by an authorized auditor, regulatory authorities or Institutional Review Boards (IRBs)

Boehringer Ingelheim's department of Quality Assurance may conduct quality control visits to the participating sites to ensure proper implementation of the study protocol and all related regulatory and BI procedures.

The Sponsor or designee (contracted CRO) will assure database quality by reviewing the data entered into the CRFs by investigational staff for completeness and accuracy, and in accordance with the data validation plan.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

The basic limitations of the study relate to the general limitations that concern non-interventional studies. Since this study is a non-interventional study, it could be possible that different parameters which were not assessed and thus remain unknown, might lead to overestimating/underestimating/non-detection of differences of specific patients' characteristics. Survival in IPF cohort studies is affected by the clinical characteristics and the related baseline patient conditions, as well as by the time interval between the diagnosis and the inclusion of the patient in the protocol. In this study, only patients with newly diagnosed IPF committed to treatment with nintedanib according to the decision of their treating physicians' will be included. This does not preclude, but definitely minimizes significant differences in the baseline characteristic of the enrolled patients.

Selection bias on the patient level will be minimized by consecutive enrollment.

No re-evaluation of patients in this study is initially foreseen, something, that can lead to the conclusion that patients with overlapping diagnoses (like fibrosing interstitial pneumonia of unknown cause) have been included in the study, thus depicting the difficulties in differential diagnosis in clinical practice. However, given the fact that the participating sites are reference centers for IPF, and considering the eligibility criteria that apply for this study, the expected bias might be low.

The study is going to provide evidence regarding the quality of life of IPF patients treated with nintedanib in reference centers that follow up about 70%-80% of IPF patients in Greece.

Given the small numbers and the heterogeneous population no comparisons and causal associations can be assessed as shown in <u>Table 3</u> in <u>Section 9.5</u>. In addition, due to the small sample size this study is rather exploratory and no definite conclusions can be drawn regarding the efficacy of nintedanib.

Regarding to patient information/recall bias that may be introduced by the collection of data pertaining to patient-reported outcomes, this will be mitigated through the use of widely used PROs that employ a short recall period as all questions refer to the symptoms and state of health at the day of completion. In addition, the self-administered PROs shall be completed by the patients themselves before the performance of any study-specific procedure(s) or clinical assessment(s) in order to avoid introducing any response bias.

#### 9.10 OTHER ASPECTS

None

## 9.10.1 Data quality assurance

Appropriate quality control procedures will be followed during this study so as to ensure quality and accuracy of the data. The delegated representative of the Sponsor (contracted CRO) will provide Investigators with a file for the archiving of all study documents. The contents of

this file may be subjected to inspection from the regulatory authorities or the Institution Review Boards (IRBs). Boehringer Ingelheim quality control department may perform audits in the participating centers in order to ensure that all study procedures are followed. The sponsor or its delegate (contracted CRO) will ensure electronic database quality through review of the captured data regarding their accuracy and completeness of data according to DMP. The eCRF data from each participating center will be saved in CD-ROM after the completion of the study and will be distributed to the centers.

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by Institutional Review Board (IRBs) /Independent Ethics Committee (IECs) or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

# 9.10.2 Study records

Case Report Forms (CRFs) for individual patients will be provided by the sponsor, either on paper or via remote data capture.

Every doctor will have a study folder containing:

- The study contract between the physician and
- The protocol
- The patient identification list (not allowed to be used off site)
- An approval letter by the Scientific Committee/Ethics Committee for the specific site
- Informed consent forms
- eCRF Sample printouts

## 9.10.2.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data reported on the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study; also, current medical records must be available.

For eCRFs all data must be derived from source documents.

#### 9.10.2.2 Direct access to source data and documents

The investigator / institution will permit study-related monitoring, audits, IRB / IEC review and regulatory inspection, providing direct access to all related source data / documents. CRFs/eCRFs and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical study monitor, auditor and inspection by health authorities (e.g. US Food and Drug Administration (FDA)). The Clinical Research Associate (CRA) / Clinical Trial Manager (CTM) and auditor may review all CRFs/eCRFs and written informed consents. The accuracy of the data will be verified by reviewing the documents described in Section 9.10.2.1.

#### 9.10.2.3 Storage of records

Patient's files and other source documents must be kept for the maximum time period permitted by the hospital/institution or as defined below. The investigator must consult with the sponsor in case they wish to transfer the files to a third party, move them to a different location or if they are not capable of maintaining them for the defined period.

The investigator should keep the study files (e.g. source documents like medical files, contracts, electronic files and signed informed consent forms) for as long as it is defined by the applicable laws and regulations. The sponsor is responsible for maintaining the documents for at least 25 years. The archived data can be kept in electronic form so long as there are available backup copies in printed form, if it is required.

The participating sites are responsible for the archiving of the necessary documents/evidence for 25 years at least or for as long as it is required by the local legislation.

# 9.10.3 Completion of study

The Institutional Review Board (Scientific/Administrative Board) in each participating hospital center needs to be notified about the end of the study (last patient out) or early termination of the study, unless it is differently required by the national regulations that govern the conduct of such studies in case these regulations have been amended until the completion of the study.

#### 10. PROTECTION OF HUMAN SUBJECTS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Tripartite Guideline for Good Clinical Practice (GCP) (to the extent applicable to the NIS setting and required by local regulations), Good Epidemiological Practice (GEP), Guidelines for Good Pharmacoepidemiology Practice (GPP), and relevant BI Standard Operating Procedures (SOPs). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol/ICH GCP.

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

# 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This study will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and Competent Authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the study, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the investigator as part of the study records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

**BI Study Number 1199-0355** 

Proprietary confidential information © 2021BoehringerIngelheim International GmbH or one or more of its affiliated companies

The patient must be informed that his/her personal study-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorized monitors (CTM/CRA) or Quality Medicine auditors appointed by Boehringer Ingelheim, by appropriate IRB / IEC members, and by inspectors from regulatory authorities.

# 10.2 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities.

Patient's private data are going to be used by Boehringer Ingelheim and will be kept according to the requirements of the EU Data Protection Directive (95/46/EC) guidelines and the 2016/679 EU regulation on the protection of natural persons with regard to the processing of personal data and on the free movement of such data and the national legislation regarding protection of private data. Data will be collected with the use of key codes. The identification codes will be used instead of patient names in order to protect patient identities when referring to study data. The level of disclosure should also be explained to the patient.

Only authorized staff (hospital staff, sponsor representatives including monitors, authority representatives) will have access to patients' private data e.g. original source documents (medical records). The patient will agree to this specifically by providing informed consent and the appropriate statement will be included in the Informed Consent Form (ICF).

The physician must comply with the confidentiality policy as it is defined within the Study Contractual Agreement. The physician will comply with the Protocol that has been approved by the Scientific Board/Ethics Committee. The physician is responsible for the conduct of all study aspects in the study site and validates the integrity of all forwarded to the sponsor data with their signature.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

#### 11.1 DEFINITIONS OF ADVERSE EVENTS

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### Adverse reaction

An adverse reaction is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse reactions may arise from use of the product within or outside the terms of the marketing authorization or from occupational exposure. Conditions of use outside the marketing authorization include off-label use, overdose, misuse, abuse and medication errors.

#### Serious adverse event

A serious adverse event is defined as any AE which

- results in death,
- is life-threatening,
- requires in-patient hospitalization, or
- prolongation of existing hospitalization,
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly/birth defect.
Life-threatening in this context refers to a reaction in which the patient was at risk of death at the time of the reaction; it does not refer to a reaction that hypothetically might have caused death if more severe.

Medical and scientific judgement should be exercised in deciding whether other situations should be considered serious reactions, such as important medical events that might not be immediately life threatening or result in death or hospitalization but might jeopardize the patient or might require intervention to prevent one of the other outcomes listed above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization or development of dependency or abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse reaction.

# Adverse Event of Special Interest (AESI)

The term Adverse Event of Special Interest (AESI) relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this study, e.g. the potential for AEs based on knowledge from other compounds in the same class.

No AESIs have been defined for this study.

# 11.2 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

The investigator shall maintain and keep detailed records of all AEs in their patient files.

## Collection of AEs

The study design is of non-interventional nature and the study is conducted within the conditions of the approved marketing authorization. Sufficient data from controlled interventional trials are available to support the evidence on the safety and efficacy of the studied BI drug. For this reason, the following AE collection and reporting requirements have been defined.

The following must be collected by the investigator in the (e)CRF from signing the informed consent onwards until the end of the study:

- all adverse drug reaction (ADRs) (serious and non-serious),
- all AEs with fatal outcome,

All ADRs, including those persisting after study completion must be followed up until they are resolved, have been sufficiently characterized, or no further information can be obtained.

The investigator carefully assesses whether an AE constitutes an ADR using the information below.

## Causal relationship of adverse event

The definition of an adverse reaction implies at least a reasonable possibility of a causal relationship between a suspected medicinal product and an adverse event. An adverse reaction, in contrast to an adverse event, is characterized by the fact that a causal relationship between a medicinal product and an occurrence is suspected.

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest a reasonable causal relationship could be:

- The event is **consistent with the known pharmacology** of the drug
- The event is known to be caused by or attributed to the drug class.
- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the **event is reproducible** when the drug is re-introduced
- No medically sound alternative etiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically **drug-related and infrequent in the general population** not exposed to drugs (e.g. Stevens-Johnson syndrome).

**BI Study Number 1199-0355** 

Proprietary confidential information © 2021BoehringerIngelheim International GmbH or one or more of its affiliated companies

• An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is diminished).

# Arguments that may suggest that there is no reasonable possibility of a causal

# Relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident
  (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days/weeks of
  drug administration; allergic reaction weeks after discontinuation of the drug
  concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives).
  - Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger.
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the study drug treatment continues or remains unchanged.

## Intensity of adverse event

The intensity of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated

Moderate: Enough discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

#### Pregnancy:

In rare cases, pregnancy might occur in a study. Once a subject has been enrolled into the study, after having taken nintedanib, the investigator must report any drug exposure during pregnancy, which occurred in a female subject or in a partner to a male subject to the Sponsor by means of Part A of the Pregnancy Monitoring Form. The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported by means of Part B of the Pregnancy Monitoring Form.

In the absence of a reportable AE, only the Pregnancy Monitoring Form must be completed, otherwise the NIS AE form is to be completed and forwarded as well within the respective timelines.

## Expedited Reporting of AEs and Drug Exposure During Pregnancy

The following must be reported by the investigator on the NIS AE form from signing the informed consent onwards until the end of the study:

| Type of Report | Timeline |
|---|---|
| All <b>serious ADRs</b> associated with Nintedanib | immediately within 24 hours |
| All <b>AEs with fatal outcome</b> in patients exposed to Nintedanib | immediately within 24 hours |
| All <b>non-serious ADRs</b> associated with Nintedanib | 7 calendar days |
| All pregnancy monitoring forms | 7 calendar days |

The same timelines apply if follow-up information becomes available for the respective events. In specific occasions the Investigator could inform the Sponsor upfront via telephone. This does not replace the requirement to complete and fax the NIS AE form.

# <u>Information required</u>

For each reportable adverse event, the investigator should provide the information requested on the appropriate (e)CRF pages and the NIS AE form.

The NIS AE form and Pregnancy Monitoring Forms should be submitted to the Pharmacovigilance Department at For details regarding

Pregnancy Monitoring Forms, please refer to <u>Section 11.2</u> paragraphs entitled, "Pregnancy" and "Expedited Reporting of AEs and Drug Exposure During Pregnancy."

## Reporting of related Adverse Events associated with any other BI drug

The investigator is encouraged to report all adverse events related to any BI drug other than the nintedanib according to the local regulatory requirements for spontaneous AE reporting at the investigator's discretion by using the locally established routes and AE report forms. The term AE includes drug exposure during pregnancy, and, regardless of whether an AE occurred or not, any abuse, off-label use, misuse, medication error, occupational exposure, lack of effect, and unexpected benefit.

#### 11.3 REPORTING TO HEALTH AUTHORITIES

Adverse event reporting to regulatory agencies will be done by the MAH according to local and international regulatory requirements.

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Participating physicians and Boehringer Ingelheim will be informed on the progress and status of the study on a regular basis. An Annual Report will be issued that contains a section on project management (recruitment status, information on technical and administrative issues) and tabular listings of data. Further, meetings of the National Scientific Committee as well as investigator meetings are planned (preferably in the context of major Pulmonology Meetings).

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

Following database lock, a final report that summarizes the tables of the analysis and explanatory text will be written by the Data Management. Data management according to our contractual agreement will prepare a final Study Report which will be used as a basis for the final Report that will be written internally. After approval from the members of the National Scientific Committee and the sponsor, a final version will be generated that may be used for regulatory purposes, but also as basis for the publications of the study.

Every effort will be made, given the collected data, in order to produce scientific publications that will in turn contribute to better care for IPF patients and justify the scientific effort. The publication strategy and the authors' list will be agreed between the Medical Department of Boehringer Ingelheim Hellas and the participating investigators. Boehringer Ingelheim Hellas will be the official owner of all collected date and results. Every study publication should be consistent with BI's publication policy and guided by the Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals of the International Committee of Medical Journals (ICMJE) (24).

This study together with the results will be posted to the web-based platform Clinicaltrials.gov (CT.gov), in the EU electronic register of post-authorization studies -ENCEPP

(www.encepp\_eu/encepp\_studies/indexRegister.shtml) and in the platform of Non-Interventional Studies (NIS) Register [Dilon (www.dilon.sfee.gr)] according to local requirements. This webpage constitutes an electronic register of the NIS conducted in Greece and is hosted as part of the Hellenic Association of Pharmaceutical Companies (SFEE) website.

#### 13. REFERENCES

## 13.1 PUBLISHED REFERENCES

- 1. Hutchinson J, Fogarty A, Hubbard R, McKeever T. Global incidence and mortality of idiopathic pulmonary fibrosis: a systematic review. The European Respiratory Journal. 2015;46(3):795-806 (R17-4824)
- 2. Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, et al. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. American Journal of Respiratory and Critical Care Medicine. 2011;183(6):788-824 (P11-07084)
- 3. Anto JM, Cullinan P. Clusters, classification and epidemiology of interstitial lung diseases: concepts, methods and critical reflections. The European Respiratory Journal Supplement. 2001;32:101s-6s (R18-2836)
- 4. Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, et al. Efficacy and Safety of Nintedanib in Idiopathic Pulmonary Fibrosis. New England Journal of Medicine. 2014;370(22):2071-82 (P14-07514)
- 5. Wilson JW, du Bois RM, King TE, Jr. Challenges in pulmonary fibrosis: 8--The need for an international registry for idiopathic pulmonary fibrosis. Thorax. 2008;63(3):285-7 (R16-3079)
- 6. Tzouvelekis A, Karampitsakos T, Kontou M, Granitsas A, Malliou I, Anagnostopoulos A, et al. Safety and efficacy of nintedanib in idiopathic pulmonary fibrosis: A real-life observational study in Greece. Pulmonary Pharmacology & Therapeutics. 2018;49:61-6 (P18-01159)
- 7. Richeldi L, Cottin V, du Bois RM, Selman M, Kimura T, Bailes Z, et al. Nintedanib in patients with idiopathic pulmonary fibrosis: Combined evidence from the TOMORROW and INPULSIS trials. Respiratory Medicine 2016.113:74-9 (P16-04370)
- 8. Kreuter M, Swigris J, Pittrow D, Geier S, Klotsche J, Prasse A, et al. Health related quality of life in patients with idiopathic pulmonary fibrosis in clinical practice: insights-IPF registry. Respiratory Research. 2017;18:139 (R17-2575)
- 9. Musellim B, Okumus G, Uzaslan E, Akgun M, Cetinkaya E, Turan O, et al. Epidemiology and distribution of interstitial lung diseases in Turkey. The Clinical Respiratory Journal. 2014;8(1):55-62 (R14-4379)
- 10. Karakatsani A, Papakosta D, Rapti A, Antoniou KM, Dimadi M, Markopoulou A, et al. Epidemiology of interstitial lung diseases in Greece. Respir Med. 2009;103(8):1122-9 (R11-5060)
- 11. Coultas DB, Zumwalt RE, Black WC, Sobonya RE. The epidemiology of interstitial lung diseases. American Journal of Respiratory and Critical Care Medicine. 1994;150(4):967-72 (R03-2075)
- 12. Gribbin J, Hubbard RB, Le Jeune I, Smith CJ, West J, Tata LJ. Incidence and mortality of idiopathic pulmonary fibrosis and sarcoidosis in the UK. Thorax. 2006;61(11):980-5 (R10-2818)
- 13. Fernandez Perez ER, Daniels CE, Schroeder DR, St Sauver J, Hartman TE, Bartholmai BJ, et al. Incidence, prevalence, and clinical course of idiopathic pulmonary fibrosis: a population-based study. Chest. 2010;137(1):129-37 (R10-2800)

- 14. Kornum JB, Christensen S, Grijota M, Pedersen L, Wogelius P, Beiderbeck A, et al. The incidence of interstitial lung disease 1995-2005: a Danish nationwide population-based study. BMC Pulmonary Medicine. 2008;8:24 (R112-0229)
- 15. Raghu G, Rochwerg B, Zhang Y, Garcia CA, Azuma A, Behr J, et al. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline: Treatment of Idiopathic Pulmonary Fibrosis. An Update of the 2011 Clinical Practice Guideline. American Journal of Respiratory and Critical Care Medicine. 2015;192(2):e3-19 (P15-07539)
- 16. Martinez FJ, Safrin S, Weycker D, et al. THe clinical course of patients with idiopathic pulmonary fibrosis. Annals of Internal Medicine. 2005;142(12\_Part\_1):963-7 (R07-0258)
- 17. Collard HR, Moore BB, Flaherty KR, Brown KK, Kaner RJ, Talmadge E. King J, et al. Acute Exacerbations of Idiopathic Pulmonary Fibrosis. American Journal of Respiratory and Critical Care Medicine. 2007;176(7):636-43 (R11-5151)
- 18. King TE, Jr., Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, et al. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. The New England Journal of Medicine. 2014;370(22):2083-92 (R14-2103)
- 19. Noble PW, Albera C, Bradford WZ, Costabel U, Glassberg MK, Kardatzke D, et al. Pirfenidone in patients with idiopathic pulmonary fibrosis (CAPACITY): two randomised trials. Lancet. 2011;377(9779):1760-9 (R11-4827)
- 20. Richeldi L, Costabel U, Selman M, Kim DS, Hansell DM, Nicholson AG, et al. Efficacy of a tyrosine kinase inhibitor in idiopathic pulmonary fibrosis. The New England Journal of Medicine. 2011;365(12):1079-87 (P11-11216)
- 21. Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, et al. Efficacy and safety of nintedanib in idiopathic pulmonary fibrosis. The New England Journal of Medicine. 2014;370(22):2071-82 (P14-07514)
- 22. Chaudhary NI, Roth GJ, Hilberg F, Muller-Quernheim J, Prasse A, Zissel G, et al. Inhibition of PDGF, VEGF and FGF signalling attenuates fibrosis. The European Respiratory Journal. 2007;29(5):976-85 (P07-07435)
- 23. Coward WR, Saini G, Jenkins G. The pathogenesis of idiopathic pulmonary fibrosis. Therapeutic Advances in Respiratory Disease. 2010;4(6):367-88 (R18-2840)
- 24. Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991;85 Suppl B:25-31; discussion 3-7 (R98-0966)
- 25. Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999;54(7):581-6 (R04-1043)
- 26. Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, et al. Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. Aids. 2002;16(4):605-13 (R18-2837)
- 27. Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Archives of Internal Medicine. 2006;166(10):1092-7 (R18-2838)
- 28. Swigris JJ, Wilson H, Esser D, Conoscenti CS, Stansen W, Kline Leidy N, et al. Psychometric properties of the St George's Respiratory Questionnaire in patients with idiopathic pulmonary fibrosis: insights from the INPULSIS trials. BMJ Open Respiratory Research. 2018;5(1):e000278 (P18-05386)
- 29. Papiris SA, Daniil ZD, Malagari K, Kapotsis GE, Sotiropoulou C, Milic-Emili J, et al. The Medical Research Council dyspnea scale in the estimation of disease severity in idiopathic pulmonary fibrosis. Respir Med. 2005;99(6):755-61 (R18-2839)

30. Manen MJG van, Birring SS, Vancheri C, Cottin V, Renzoni EA, Russell A-M, et al. Cough in idiopathic pulmonary fibrosis. European Respiratory Review. 2016;25(141):278-86 (P18-00823)

# 13.2 UNPUBLISHED REFERENCES

*Not applicable* 

c25576073-03

Proprietary confidential information © 2021BoehringerIngelheim International GmbH or one or more of its affiliated companies

# ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

Not applicable

# ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

| Study title: Investigating Trends in Quality of Life in Patients with IPF Under Treatment | | | | | |
|---|---|---|---|---|---|
| Stat | with Nintedanib | iiCiiiS W | <i>,,,,</i> | Onaci | 11 Catiment |
| | win Nimedanio | | | | |
| Stuc | ly reference number: | | | | |
| Sect | ion 1: Milestones | Yes | No | N/A | Section |
| | | | | | Number |
| 1.1 | Does the protocol specify timelines for | | | | |
| | 1.1.1 Start of data collection | | | | 6 |
| | 1.1.2 End of data collection | | | | 6 |
| | 1.1.3 Study progress report(s) | | | | |
| | 1.1.4 Interim progress report(s) | | | | |
| | 1.1.5 Registration in the EU PAS register | | | | |
| | 1.1.6 Final report of study results. | | | | 6 |
| Comr | nents: | | I | | |
| 1.1.3 | S → Not required according to national requirements | for non | -interv | ventiona | al studies |
| 1.1.4 | → Not required as no interim analysis of data is sch | eduled | | | |
| 1.1.5 | 5 → The present study has not yet been registered | in the I | Europe | an Unio | on electronic |
| Regi | ster of Post-Authorisation Studies (EU PAS register) | ). | | | |

| Secti | on 2: Research question | Yes | No | N/A | Section |
|---|---|---|---|---|---|
| | | | | | Number |
| 2.1 | Does the formulation of the research question and | | | | |
| | objectives clearly explain: | | | | |
| | 2.1.1 Why the study is conducted? (e.g. to | | | | |
| | address an important public health concern, a | | | | 8 |
| | risk identified in the risk management plan, an | | | | |
| | emerging safety issue) | | | | |
| | 2.1.2 The objective(s) of the study? | | | | 8 |
| | 2.1.3 The target population? (i.e. population or | | | | |
| | subgroup to whom the study results are | | | | 9.2.2 |
| | intended to be generalized) | | | | |
| | 2.1.4 Which hypothesis(-es) is (are) to be tested? | | | | |
| | 2.1.5 If applicable, that there is no <i>a priori</i> | | | | |
| | hypothesis? | | Ш | | |
| Comn | nents: | | | | |
| 2.1.4 | & 2.1.5 $\rightarrow$ No hypothesis testing is going to be perfo | ormed t | herefor | e no sp | ecific effects |
| or en | dpoints are defined. | | | | |
| Secti | on 3: Study design | Yes | No | N/A | Section |
| | | | | | Number |
| 3.1 | Is the study design described? (e.g. cohort, case- | | | | |
| | control, cross-sectional, new or alternative | | | | 9.1 |
| | design) | | | | |
| 3.2 | Does the protocol specify whether the study is | | | | |
| | based on primary, secondary or combined data | $\boxtimes$ | | | 9.4 |
| | collection? | | | | |

| Secti | etion 3: Study design | | No | N/A | Section |
|---|---|---|---|---|---|
| | | | | | Number |
| 3.3 | Does the protocol specify measures of | $\boxtimes$ | | | 9.4 |
| | occurrence? (e.g. incidence rate, absolute risk) | | | | 9.4 |
| 3.4 | Does the protocol specify measure(s) of | | | | |
| | association? (e.g. relative risk, odds ratio, excess | | $\boxtimes$ | | |
| | risk, incidence rate ratio, hazard ratio, number | | | | |
| | needed to harm (NNH) per year) | | | | |
| 3.5 | Does the protocol describe the approach for the | | | | |
| | collection and reporting of adverse events/adverse | $\bowtie$ | | | 11 |
| | reactions? (e.g. adverse events that will not be | | | | 11 |
| | collected in case of primary data collection) | | | | |
| Comn | nents: | | | | |
| Secti | on 4: Source and study populations | Yes | No | N/A | Section |
| | | | | | Number |
| 4.1 | Is the source population described? | | | | 9.1 |
| 4.2 | Is the planned study population defined in terms | | | | 9.2.2 |
| | of: | | | | 9.2.2 |
| | 4.2.1 Study time period? | | | | |
| | 4.2.2 Age and sex? | | | | |
| | 4.2.3 Country of origin? | | | | |
| | 4.2.4 Disease/indication? | | | | 9.2.2 |
| | 4.2.5 Duration of follow-up? | | | | |

| Sect | ion 4: Source and study populations | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 4.3 | Does the protocol define how the study population will be sampled from the source population? (e.g. event or inclusion/exclusion criteria) | | | | 9.2.2 |
| Comn | nents: | | | | |
| Sect | ion 5: Exposure definition and measurement | Yes | No | N/A | Section<br>Number |
| 5.1 | Does the protocol describe how the study exposure is defined and measured? (e.g. operational details for defining and categorising exposure, measurement of dose and duration of drug exposure) | | | | 9.3.1 |
| 5.2 | Does the protocol address the validity of the exposure measurement? (e.g. precision, accuracy, use of validation sub-study) | $\boxtimes$ | | | 9.3.1 |
| 5.3 | Is exposure classified according to time windows? (e.g. current user, former user, non-use) | | | | |
| 5.4 | Is exposure classified based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | | | |
| Comn | nents: | • | | | |
| 5.2. | This is new data collection, thus the accuracy of expo | osure in | format | ion is ve | ery high |

| Sect | ion 6: Outcome definition and measurement | Yes | No | N/A | Section |
|---|---|---|---|---|---|
| | | | | | Number |
| 6.1 | Does the protocol specify the primary and secondary (if applicable) outcome(s) to be investigated? | | | | 9.3.2 |
| 6.2 | Does the protocol describe how the outcomes are defined and measured? | | | | 9.3.2 |
| 6.3 | Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, prospective or retrospective ascertainment, use of validation sub-study) | | | | 9.5 |
| 6.4 | Does the protocol describe specific endpoints relevant for Health Technology Assessment? (e.g. HRQoL, QALYs, DALYS, health care services utilisation, burden of disease, disease management) | | | | 9.3.2 |
| Comn | nents | | | | |
| Sect | ion 7: Bias | Yes | No | N/A | Section<br>Number |
| 7.1 | Does the protocol describe how confounding will be addressed in the study? | | | $\boxtimes$ | |
| | 7.1.1. Does the protocol address confounding by indication if applicable? | | | $\boxtimes$ | |
| 7.2 | Does the protocol address: | | | | |
| | 7.2.1. Selection biases (e.g. healthy user bias) | | | | 9.2.2 |

| Sect | ion 7: Bias | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| | 7.2.2. Information biases (e.g. misclassification of exposure and endpoints, time-related bias) | $\boxtimes$ | | | 9.2.2 |
| 7.3 | Does the protocol address the validity of the study covariates? | | | $\boxtimes$ | |
| Comn | nents: | | | | |
| No confounders or effect modifiers are discussed since no hypothesis testing or assessment of effects is being performed. | | | | | |
| Sect | ion 8: Effect modification | Yes | No | N/A | Section<br>Number |
| 8.1 | Does the protocol address effect modifiers? (e.g. collection of data on known effect modifiers, sub-group analyses, anticipated direction of effect) | | | | |
| Comn | nents: | | | | |
| Sect | ion 9: Data sources | Yes | No | N/A | Section<br>Number |
| 9.1 | Does the protocol describe the data source(s) used in the study for the ascertainment of: | | | | |
| | 9.1.1 Exposure? (e.g. pharmacy dispensing, general practice prescribing, claims data, self-report, face-to-face interview) | $\boxtimes$ | | | 9.3.1, 9.4 |

| Sect | ion 9: Data sources | Yes | No | N/A | Section |
|---|---|---|---|---|---|
| | | | | | Number |
| | 9.1.2 Outcomes? (e.g. clinical records, laboratory markers or values, claims data, self-report, patient interview including scales and questionnaires, vital statistics) | | | | 9.3.2, 9.4 |
| | 9.1.3 Covariates? | | | | 9.3.3, 9.4 |
| 9.2 | Does the protocol describe the information available from the data source(s) on: | | | | |
| | 9.2.1 Exposure?(e.g. date of dispensing, drug quantity, dose, number of days of supply prescription, daily dosage, prescriber) | | | | 9.4 |
| | 9.2.2 Outcomes?(e.g. date of occurrence, multiple event, severity measures related to event) | $\boxtimes$ | | | 9.4 |
| | 9.2.3 Covariates? (e.g. age, sex, clinical and drug use history, co-morbidity, co-medications, lifestyle) | | | | 9.4 |
| 9.3 | Is a coding system described for: | | | | |
| | 9.3.1 Exposure? (e.g. WHO Drug Dictionary, Anatomical Therapeutic Chemical (ATC) Classification System) | | | | |
| | 9.3.2 Outcomes?(e.g. International Classification of Diseases (ICD)-10, Medical Dictionary for Regulatory Activities (MedDRA)) | | $\boxtimes$ | | |
| | 9.3.3 Covariates? | | | | |
| 9.4 | Is a linkage method between data sources described?(e.g. based on a unique identifier or other) | $\boxtimes$ | | | 9.4 |

| Comm | nents: | | | | |
|---|---|---|---|---|---|
| Secti | on 10: Analysis plan | Yes | No | N/A | Section<br>Number |
| 10.1 | Is the choice of statistical techniques described? | | | | 9.7.1 |
| 10.2 | Are descriptive analyses included? | | | | 9.5 |
| 10.3 | Are stratified analyses included? | | | | |
| 10.4 | Does the plan describe methods for adjusting for confounding? | | | | |
| 10.5 | Does the plan describe methods for handling missing data? | | | | 9.7.1 |
| 10.6 | Is sample size and/or statistical power estimated? | | | | 9.5 |
| Comm | nents: | l | | | |
| <u>Secti</u> | on 11: Data management and quality control | Yes | No | N/A | Section<br>Number |
| 11.1 | Does the protocol provide information on data<br>storage?(e.g. software and IT environment,<br>database maintenance and anti-fraud protection,<br>archiving) | $\boxtimes$ | | | 9.8, 9.10.2 |
| 11.2 | Are methods of quality assurance described? | | | | 9.8 |
| 11.3 | Is there a system in place for independent review of study results? | | | | |
| Comm | nents: | | | | |
| 11.3- | → The study design does not require an independent | review | of the | results. | |

| Section 12: Limitations Yes No N/A Section Number 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical | |
|---|---|
| Number | |
| Number | |
| 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical | l |
| results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical | r |
| 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical | |
| 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical | |
| 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical | |
| (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical | |
| such biases, validation sub-study, use of validation and external data, analytical | |
| validation and external data, analytical | |
| 4112 | |
| methods) | |
| 12.2 Does the protocol discuss study feasibility? | |
| (e.g. study size, anticipated exposure, duration of | |
| follow-up in a cohort study, patient recruitment) | |
| Comments: | |
| Section 13: Ethical issues Yes No N/A Section | l |
| Number | r |
| 13.1 Have requirements of Ethics Committee/ | |
| Institutional Review Board been described? | |
| 13.2 Has any outcome of an ethical review procedure | |
| been addressed? | _ |
| 13.3 Have data protection requirements been | |
| described? | |

| Comments: | | | | |
|---|---|---|---|---|
| Section 14: Amendments and deviations | Yes | No | N/A | Section<br>Number |
| 14.1 Does the protocol include a section to document amendments and deviations? | | | | 5 |
| Comments: | • | l | | |
| Section 15: Plans for communication of study results | Yes | No | N/A | Section |
| | | | | Number |
| 15.1 Are plans described for communicating study results (e.g. to regulatory authorities)? | $\boxtimes$ | | | 12 |
| 15.2 Are plans described for disseminating study results externally, including publication? | | | | 12 |
| Comments: | 1 | | , | |

# **ANNEX 3. ADDITIONAL INFORMATION**

# ST. GEORGE'S RESPIRATORY QUESTIONNAIRE (SGRQ)

This questionnaire is designed to help us learn much more about how your breathing is troubling you and how it affects your life. We are using it to find out which aspects of your illness cause you most problems, rather than what the doctors and nurses think your problems are.

Please read the instructions carefully and ask if you do not understand anything. Do not spend too long deciding about your answers.

| Before completing the rest of the questionnaire: | | | | | |
|---|---|---|---|---|---|
| Please tick in one box to show how you describe your current health: | Very good | Good | Fair | Poor | Very<br>poor |
| Copyright reserved | | | | | |
| | | | Tel.<br>Fax | | |

## **UK/** English (original) version

 $f:\label{limit} f:\label{limit} f:\label{lim$ 

# St. George's Respiratory Questionnaire, Continued 

## PART 1

| Questi | ions about how much chest trouble you have | had over | the past | 4 weeks. | | |
|---|---|---|---|---|---|---|
| | | Ple | ase tick (✔ | ) one box | for each qu | estion: |
| | | most<br>days<br>a week | several<br>days<br>a week | a few<br>days<br>a month | only with<br>chest<br>infections | not<br>at<br>all |
| 1. | Over the past 4 weeks, I have coughed: | | | | | |
| 2. | Over the past 4 weeks, I have brought up phlegm (sputum): | | | | | |
| 3. | Over the past 4 weeks, I have had shortness of breath: | | | | | |
| 4. | Over the past 4 weeks, I have had attacks of wheezing: | | | | | |
| 5. | During the past 4 weeks, how many severe or vunpleasant attacks of chest trouble have you have | • | | 51 | | |
| | | | more the | Ple<br>an 3 attacl | ease tick (✔) | ) one: |
| | | | more un | an 3 attack<br>3 attack | | |
| | | | | 2 attack | | |
| | | | | 1 attac | | |
| | | | | no attacl | | |
| 6. | How long did the worst attack of chest trouble la<br>(Go to question 7 if you had no severe attacks) | | | | | |
| | (00.00 44000000 1 11 900 1100 110 001 010 0110010) | | | Ple | ease tick (✔) | ) one: |
| | | | a w | eek or mo | re 📙 | |
| | | | 3 о | r more day | /s | |
| | | | | 1 or 2 day | ys 📙 | |
| | | | less | s than a da | ау 📙 | |
| 7. | Over the past 4 weeks, in an average week, ho (with little chest trouble) have you had? | w many go | ood days | | | |
| | (with fittle chest trouble) have you had: | | | Ple | ease tick (✔) | ) one: |
| | | | No | good day | ys $\square$ | |
| | | | 1 or 2 | 2 good day | /s 🗌 | |
| | | | 3 or 4 | 4 good day | /s 🗌 | |
| | | ne | arly every | day is goo | od 🗌 | |
| | | | every | day is goo | od 🗌 | |
| 8. | If you have a wheeze, is it worse in the morning | g? | | | , | |
| | | | | | ease tick (✔) | ) one: |
| | | | | | lo 📙 | |
| | | | | Yε | es 📖 | |

# St. George's Respiratory Questionnaire, Continued 

# PART 2

| Section 1 | | | |
|---|---|---|---|
| Section 1 | | | |
| How would you describe your chest condition? | | Discos | #:-!- ( <b>/</b> ) |
| The me | oot impo | | e tick (✔) one: |
| | | rtant problem I have | |
| Cause | • | ite a lot of problems | |
| | | me a few problems | |
| | | Causes no problem | |
| If you have ever had paid employment. | | | |
| | | | e tick (✓) one: |
| • | | stop work altogether | |
| | My chest trouble interferes with my work or made me change my work | | |
| My chest trou | uble doe | s not affect my work | |
| Section 2 | | | |
| Questions about what activities usually make you fe | eel breat | hless <u>these days</u> . | |
| | | n <b>each box</b> that<br>ou <b>these days</b> : | |
| | True | False | |
| Sitting or lying still | | | |
| Getting washed or dressed | | | |
| Walking around the home | | | |
| Walking outside on the level | | | |
| Walking up a flight of stairs | | | |
| Walking up hills | | | |
| Playing sports or games | | | |

# St. George's Respiratory Questionnaire, Continued 

| PART 2 | | | | |
|---|---|---|---|---|
| Section 3 | | | | |
| Some more questions about your cough and breath | lessness | these day | <u>s</u> . | |
| | | in <b>each bo</b><br>ou <b>these da</b> | | |
| My cough hurts My cough makes me tired I am breathless when I talk I am breathless when I bend over My cough or breathing disturbs my sleep I get exhausted easily | True | False | | |
| Section 4 | | | | |
| Questions about other effects that your chest troub | le may ha | ave on you | these da | <u>ys</u> . |
| | | | | ach box that<br>these days: |
| | | | True | False |
| My cough or breathing is emb | arrassing | in public | | |
| My chest trouble is a nuisance to my family, frie | nds or ne | ighbours | | |
| l get afraid or panic when I car | not get m | ny breath | | |
| I feel that I am not in control of | my chest | problem | | |
| I do not expect my ches | st to get a | ny better | | |
| I have become frail or an invalid be | cause of | my chest | | |
| | is not sa | - | | |
| Everything seems too | much of | an effort | | |
| Section 5 | | | | |
| Questions about your medication, if you are receiving to section 6. | ng no me | edication go | o straight | |
| | | in <b>each bo</b><br>u <b>these da</b> | | |
| | True | False | | |
| My medication does not help me very much | | | | |
| I get embarrassed using my medication in public | | | | |
| I have unpleasant side effects from my medication | | | | |
| My medication interferes with my life a lot | | | | |

# St. George's Respiratory Questionnaire, Continued 

# PART 2

Section 6

These are questions about how your activities might be affected by your breathing.

| | | ck (✓) in <b>each</b> | | |
|---|---|---|---|---|
| | | you <b>because</b> | True | False |
| I take a long time to ge | et washed | l or dressed | | |
| I cannot take a bath or shower | | | | |
| I walk slower than other peop | | Ü | | |
| Jobs such as housework take a long time, or l | | - | | |
| _ | | • | | |
| If I walk up one flight of stairs, I have | • | | | |
| If I hurry or walk fast, I have | • | | | |
| My breathing makes it difficult to do things such as walk up up stairs, light gardening such as weeding, dance, p | | , , , | | |
| My breathing makes it difficult to do things such as carry garden or shovel snow, jog or walk at 5 miles per hou | • | • | | |
| My breathing makes it difficult to do things such as very run, cycle, swim fast or pla | | | | |
| Section 7 | | | | |
| We would like to know how your chest <u>usually</u> affect | ts your d | aily life. | | |
| | | ch box that ap | | |
| you beca | True | False | ubie. | |
| I cannot play sports or games | | | | |
| I cannot go out for entertainment or recreation | | | | |
| I cannot go out of the house to do the shopping | | | | |
| I cannot do housework | | | | |
| I cannot move far from my bed or chair | | | | |

# St. George's Respiratory Questionnaire, Continued 

| Here is a list of other activities that your chest trouble may prevent you doing. (You do not have to tick hese, they are just to remind you of ways in which your breathlessness may affect you): |
|---|
| Going for walks or walking the dog |
| Doing things at home or in the garden |
| Sexual intercourse |
| Going out to church, pub, club or place of entertainment |
| Going out in bad weather or into smoky rooms |
| Visiting family or friends or playing with children |
| Please write in any other important activities that your chest trouble may stop you |
| doing: |
| Now would you tick in the box (one only) which you think best describes how your chest affects you: |
| It does not stop me doing anything I would like to do $\Box$ |
| It stops me doing one or two things I would like to do $\Box$ |
| It stops me doing most of the things I would like to do $\Box$ |
| It stops me doing everything I would like to do $\Box$ |
| Thank you for filling in this questionnaire. Before you finish would you please check to see that you have answered all the questions. |

# Modified Medical Research Council (mMRC) Dyspnea Scale

#### **Grade**

- 0 "I only get breathless with strenuous exercise"
- 1 "I get short of breath when hurrying on the level or walking up a slight hill"
- 2 "I walk slower than people of the same age on the level because of breathlessness, or I have to stop for breath when walking on my own pace on the level"
- 3 "I stop for breath after walking about 100 yards or after a few minutes on the level"
- 4 "I am too breathless to leave the house" or "I am breathless when dressing"

NB: This is the modified MRC scale that uses the same descriptors as the original MRC scale in which the descriptors are numbered 1-5. The modified MRC scale (0-4) is used for calculation of BODE index.

# Cough - Visual Analogue Scale (Cough - VAS) Patient's Assessment of Cough VAS

How much cough have you had because of your idiopathic pulmonary fibrosis (IPF) in the past week?

Place a vertical ( ) mark on the line to indicate the intensity of the cough.

| No cough | Moderate cough | Intense cough |
|----------|----------------|---------------|
| 0 | 50 | 100 |
| 0 | | 100 |

# Simplified Medication Adherence Questionnaire (SMAQ) 1

Adapted for the treatment of idiopathic pulmonary fibrosis (IPF)

| 1. | Do you | u ever forget to take your medication for IPF? | YES |
|---|---|---|---|
| | | | NO |
| 2. | Do you | u always take your medication for IPF at the indicated | YES |
| | time? | | NO |
| 3. | Somet | times if you feel worse, do you stop taking your | YES |
| | medic | ation for IPF? | NO |
| 4. | Did yo | u miss your medication for IPF last weekend? | YES |
| | | | NO |
| 5. | Think | on the last week. | A: Never |
| | How o | ften did you miss your medication for IPF? | B: 1 - 2 |
| | | | C: 3 - 5 |
| | | | D: 6 - 10<br>E: More than 10 |
| | | | E. More than 10 |
| 6. | Think o | n the past 3 months. | |
| | a) | How many days have you missed your medication for IPF? | Days |
| | b) | How many days have you missed one of the two daily doses of your medication for IPF? | Days |

Adapted from (1) Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, Kindelan JM, Carmona A, Juega J, Ocampo A; on behalf of the GEEMA Study Group. AIDS 2002;16(4):605-13.

c25576073-03

Proprietary confidential information © 2021BoehringerIngelheim International GmbH or one or more of its affiliated companies

SMAK - United States/English / Mapi. SMAQ\_TS1.0\_eng-USori.doc

# Simplified Medication Adherence Questionnaire (SMAQ) <sup>1</sup>, Continued (Page 2 of 2)

The patient is considered non-adherent if:

- 1: YES
- 2: NO
- **3: YES**
- 4: YES
- 5: C, D or E
- 6: a) More than two (2) days
  - b) More than four (4) days

The questionnaire is dichotomic, any answer in the sense of non-adherent is considered non-adherent.

You can use the question number 5 as semi-quantitative:

A: 95 - 100% compliance

B: 85-94% C: 65-84% D: 30-64% E: < 30%

Adapted from (1) Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, Kindelan JM, Carmona A, Juega J, Ocampo A; on behalf of the GEEMA Study Group. AIDS 2002;16(4):605-13.

SMAK - United States/English / Mapi. SMAQ TS1.0\_eng-USori.doc

# **GAD - 7**

| GAD-7 | | | | |
|---|---|---|---|---|
| Over the last 2 weeks, how often have you been bothered by the following problems? (Use ** to indicate your answer) | Not<br>at all | Several<br>days | More than<br>half the<br>days | Nearly<br>every day |
| Feeling nervous, anxious or on edge | 0 | 1 | 2 | 3 |
| 2. Not being able to stop or control worrying | 0 | 1 | 2 | 3 |
| 3. Worrying too much about different things | 0 | 1 | 2 | 3 |
| 4. Trouble relaxing | 0 | 1 | 2 | 3 |
| 5. Being so restless that it is hard to sit still | 0 | 1 | 2 | 3 |
| Becoming easily annoyed or irritable | 0 | 1 | 2 | 3 |
| Feeling afraid as if something awful<br>might happen | 0 | 1 | 2 | 3 |

(For office coding: Total Score T\_\_\_ = \_\_ + \_\_\_ + \_\_\_)

Developed by Drs. Robert L. Spitzer, Janet B.W. Williams, Kurt Kroenke and colleagues, with an educational grant from Pfizer Inc. No permission required to reproduce, translate, display or distribute.